

#### CLINICAL STUDY PROTOCOL

# A 52-Week Open-Label Extension Study of Pimavanserin in Children and Adolescents with Irritability Associated with Autism Spectrum Disorder (ASD)

**Protocol Number:** ACP-103-070

**Amendment 3-Consolidated** 

**EudraCT Number: 2021-005388-32** 

EUCT Number: 2024-512202-25-00

ClinicalTrials.gov Number: NCT05555615

Original Protocol Date: 30 April 2021

Protocol Amendment 1 Date: 07 December 2021

**Protocol Amendment 2 Date:** 25 March 2022

Protocol Amendment 3 Date: 21 December 2022

**Protocol Amendment 3-IT Date:** 12 July 2023

Protocol Amendment 3-Consolidated Date: 29 February 2024

Protocol Template Version: 0.2

#### **Confidentiality Statement**

This protocol is the confidential information of Acadia Pharmaceuticals Inc. and is intended solely for the guidance of the clinical investigation. This protocol may not be disclosed to parties not associated with the clinical investigation or used for any purpose without the prior written consent of Acadia Pharmaceuticals Inc.

## **SPONSOR SIGNATURE PAGE**

**Title:** A 52-Week Open-Label Extension Study of Pimavanserin in Children and Adolescents with Irritability Associated with Autism Spectrum Disorder (ASD)



Final Version: 2.0

# Signature Page for ACP-103-070 OLE Protocol Amendment 3 - Consolidated

| Approve | PPD |
|---------|-------------------------------|
| | 14-Mar-2024 17:18:01 GMT+0000 |
| Approve | PPD |
| | 14-Mar-2024 17:21:43 GMT+0000 |

Signature Page for ACP-103-070 OLE Protocol Amendment 3 - Consolidated

Study: ACP-103-070 Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

## **DECLARATION OF INVESTIGATOR**

I confirm that I have read the above protocol. I understand it, and I will work according to the moral, ethical, and scientific principles governing clinical research as set out in the principles of Good Clinical Practice, as required by International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Guideline E6 and as described in the United States (US) Code of Federal Regulations (CFR) 21 CFR parts 50, 54, 56, 312, and according to applicable local requirements.

## **Confidentiality Statement**

The confidential information in this document is provided to you as an Investigator or Consultant for review by you, your staff, and the applicable institutional review board/ethics committee. Your acceptance of this document constitutes agreement that you will not disclose the information contained herein to others without written authorization from the Sponsor.

| Investigator | |
|----------------|------|
| Signature | Date |
| Name (printed) | |

# PROTOCOL SYNOPSIS

| Protocol number | ACP-103-070 Pediatric OLE |
|---|---|
| Protocol title | A 52-Week Open-Label Extension Study of<br>Pimavanserin in Children and Adolescents with<br>Irritability Associated with Autism Spectrum<br>Disorder (ASD) |
| Name of investigational product | Pimavanserin (capsules) |
| Indication | Irritability associated with ASD |
| Phase of development | 2 |
| Sponsor | Acadia Pharmaceuticals Inc.<br>12830 El Camino Real, Suite 400<br>San Diego, CA 92130 USA |
| Safety hypothesis | Pimavanserin, a selective serotonin receptor (5-HT <sub>2A</sub> ) inverse agonist/antagonist will be a safe and well tolerated treatment for children and adolescents with ASD. |
| Primary objective | Primary endpoints |
| To evaluate the long-term safety and tolerability of pimavanserin after 52 weeks of treatment in children and adolescents with ASD | <ul> <li>Treatment-emergent adverse events (TEAEs)</li> <li>Safety will also be evaluated by analyses of the following: <ul> <li>Vital signs</li> <li>Weight and body mass index (BMI)</li> <li>12-lead electrocardiograms (ECGs)</li> <li>Physical examination results</li> <li>Clinical laboratory tests (including urinalysis) and hormonal assessments</li> <li>Columbia—Suicide Severity Rating Scale (C-SSRS)</li> <li>Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A)</li> </ul> </li> </ul> |
| Efficacy hypothesis | Pimavanserin, a selective 5-HT <sub>2A</sub> inverse agonist/antagonist, will be effective in the treatment of ASD symptoms. |


#### Secondary objective Secondary endpoint To evaluate the continued Proportion of subjects who have at least 25% reduction in the Aberrant Behavior response to long-term pimavanserin treatment in Checklist-Irritability (ABC-I) subscale score children and adolescents with AND a Clinical Global Impression-Improvement (CGI-I) of irritability ASD score of 1 (very much improved) or 2 (much improved) compared to the antecedent study baseline status at Week 52 **Exploratory objectives Exploratory endpoints** To evaluate the continued Change from Baseline at Week 52 in the benefit of long-term caregiver-rated ABC subscale scores: pimavanserin treatment on the o Irritability symptoms of ASD, in children and adolescents with ASD in Stereotypic behavior the following clinical areas: Lethargy Aberrant Behavior Hyperactivity Checklist (ABC) o Inappropriate speech symptom domains Change from Baseline at Week 52 in the Maintenance of benefit Clinical Global Impression—Severity (CGI-S) Response to treatment of irritability score CGI-I of irritability score from antecedent study Baseline at Week 52 Change from Baseline at Week 52 in the Caregiver Strain Questionnaire (CGSQ) Proportion of subjects who have at least 25% reduction from the antecedent study Baseline in the ABC-I subscale score (ABC-I responders) at Week 52 Proportion of subjects who have CGI-I of irritability score of 1 (very much improved) or 2 (much improved) compared to the antecedent study baseline status (CGI-I of irritability responders) at Week 52 **Number of study sites** Approximately 60 global sites and approximately eight countries will participate in this study.

| Number of subjects planned | The planned sample size is not based on statistical power but will depend on the number of subjects who complete the antecedent double-blind study and who rollover into this open-label extension (OLE) study. |
|---|---|
| Test product, dose, and administration | Pimavanserin "low dose" (see below details), or pimavanserin "high dose" (see below details), administered orally, once daily. |
| | <u>Dose</u> |
| | Subjects will be stratified by age group (5- through 12-year-olds or 13- through 17-year-olds). Subjects will remain in the age group they were stratified into during the antecedent double-blind study, throughout the OLE study. |
| | Each age group has its own "low dose" and high dose". For the 5- through 12-year-olds, the "low dose" will be 10 mg/day pimavanserin, and the "high dose" will be 20 mg/day pimavanserin. For the 13- through 17-year-olds, the "low dose" will be 20 mg/day pimavanserin and the "high dose" will be 34 mg/day pimavanserin. |
| | All subjects will receive once daily (QD) doses of pimavanserin over 52 weeks of treatment. |
| | Within each age group, eligible subjects will receive pimavanserin "low dose" for the first two weeks of the study. At the Week 2 visit, the dose may be increased to pimavanserin "high dose", based on the Investigator's assessment of clinical response. |
| | After the Week 2 visit, and up to and including the Week 20 visit, dose adjustments, either increases or decreases, may be made at any clinic visit (scheduled or unscheduled), based on the Investigator's assessment of clinical response and tolerability. |
| | No further dose adjustments are allowed after the Week 20 visit. |
| | Pimavanserin dosages below: Pimavanserin 10 mg (provided as 1×10 mg capsule) |
| | Pimavanserin 20 mg (provided as 1×20 mg capsule) |
| | Pimavanserin 34 mg (provided as 1×34 mg capsule) |
| Study design | This study will be conducted as a 52-week, open-label extension study of the antecedent double-blind study |

to determine the long-term safety and tolerability of pimavanserin for the treatment of irritability associated with ASD in children and adolescents (5 through 17 years old at the time of enrolling into the antecedent double-blind study).


Date: 29 February 2024

Subjects who have completed the antecedent double-blind study and who have shown no significant worsening of symptoms at the end of the study as evidenced by the CGI-I of irritability will be included in this long-term extension study.

Study ACP-103-070 subjects must be consented prior to the procedures being performed at the End of Treatment (EOT) visit in the antecedent double-blind study. Procedures performed at the EOT visit of the antecedent double-blind study will be carried over to the ACP-103-070 study to be included as baseline information, and this visit will be considered the Baseline Visit (Visit 1) of the ACP-103-070 study.

An independent data and safety monitoring board (DSMB) will review interim safety data including data on TEAEs and serious TEAEs.

The study will have two periods:

- Open-label treatment period (52 weeks)
- Safety follow-up period (at least 30 days)

The study design schema is provided in Figure S–1. The schedule of assessments is provided in Table S-1.

#### **Open-Label Treatment Period (52 weeks)**

During the treatment period, clinic visits will be conducted at Baseline and Weeks 2, 6, 12, 20, 28, 36, 44, and 52, or upon early termination (ET) from the study.

Study drug will be dispensed to the subject to take home at the Baseline visit and at each subsequent clinic visit. The subject and their parent/legally acceptable representative (LAR) will be provided instructions for the subject's first dose of study drug the day after the Baseline visit. It is recommended that the subject take the study drug at approximately the same time each day as a single, oral dose.

All concomitant medications should remain at a stable dose throughout the study, if possible, except as

| | T |
|---|---|
| | described in Appendix A to minimize confounding interpretation of any correlating pimavanserin dose changes, including treatment discontinuations. |
| | Safety Follow-up Period (30[+3] days) |
| | A follow-up safety assessment will be conducted by telephone call at least 30 days after the last dose of study drug. |
| Study duration | The duration of participation for individual study subjects will be up to approximately 56 weeks, consisting of a 52-week open-label treatment period, and a safety follow-up period of at least 30(+3) days (Figure S-1). |
| | The study start date is defined as the date the first subject is enrolled, which is the Baseline visit date the first subject for this open-label study. |
| | The primary completion date is the last date that subject data was collected for the primary outcome measure. |
| | The study completion date (End of Study) is defined as the last date that subject data was collected, which includes the safety follow-up telephone call visit. The total duration of exposure to pimavanserin may be greater than 52 weeks (e.g., up to 58 weeks) as some subjects have been treated with pimavanserin in an antecedent double-blind study. |
| Main criteria for inclusion and exclusion | To be eligible for this study, subjects must meet all of<br>the inclusion criteria and none of the exclusion criteria<br>to enter this open-label extension study. |
| | Inclusion Criteria: |
| | Study Population |
| | Has completed the treatment period of the antecedent double-blind study |
| | 2. Informed consent prior to the conduct of any study procedures is required as follows: |
| | a. The subject should provide written or oral assent if deemed able by the Investigator. |

b. The subject's parent/LAR must provide written consent. The subject's parent/LAR must be considered reliable by the Investigator, able to complete assessments regarding the subject's development and behavior throughout the study, and able to help ensure compliance with study treatment, study visits, and protocol procedures


Date: 29 February 2024

c. If a person other than the parent/LAR has been designated as a caregiver for the purpose of providing input for caregiver-reported scales, that person must also provide written consent. Such a designee should be a family member, adult and responsible, living with or in very frequent contact with the subject participating in the study, who is committed to providing responses for the caregiver-reported scales for the duration of the study

The process of obtaining informed consent will be conducted in accordance with institutional review board (IRB) or ethics committee (EC) policy and applicable local law.

3. In the Investigator's opinion, the subject, to the best of his/her ability, the parent/LAR, and the designated caregiver (if applicable, and in accordance with IRB or EC policy and applicable local law) are able to understand the nature of the study, follow protocol requirements and be willing to comply with study drug administration requirements

#### Psychiatric Diagnosis

- 4. Continues to be both clinically stable and not at imminent risk of suicide or injury to self, others, or property, in the opinion of the Investigator
- 5. Continues to be medically stable at enrollment, in the opinion of the Investigator

#### **Contraceptives**

6. Female subjects who participate in this study must either be unable to become pregnant (e.g., premenarchal, surgically sterile, etc.) -OR- must agree to use two clinically acceptable methods of contraception (e.g., oral, intrauterine device [IUD], diaphragm plus spermicide, injectable, transdermal or implantable contraception) during the treatment period, and for at least 45 days after last dose.

Final Version: 2.0 Date: 29 February 2024

All female subjects of childbearing potential must have a negative urine human chorionic gonadotropin (hCG) pregnancy test at Baseline and all clinic visits. Females of childbearing potential are defined as females who have begun menstruating.

#### **Exclusion Criteria:**

#### Study Population

1. Subject or parent/LAR is judged by the Investigator to be inappropriate for the study (e.g., significantly noncompliant in the antecedent double-blind study)

## CNS, Psychiatric, and Illicit Drug Use Criteria

- 2. Requires treatment with a medication prohibited by the protocol, including concomitant psychotropic drugs targeting irritability, including those used off-label (clonidine, guanfacine, and propranolol; lithium, valproate), medications that prolong the QT interval; and strong cytochrome P450 (CYP) 3A4 enzyme (CYP3A4) inhibitors and inducers (see Appendix A and Appendix B)
- 3. Is at a significant risk of suicide, or is a danger to self or others, in the opinion of the Investigator based upon all available sources of information including C-SSRS (positive answer to suicidal ideation questions 4 or 5 [or positive answer to suicidal behavior questions at Baseline])
- 4. Is at risk of significant violent behavior to the extent that participation would pose an undue

risk to other patients, caregivers, or others in the opinion of the Investigator


Date: 29 February 2024

5. Has a positive urine drug test at Baseline. For study eligibility, the urine toxicology (drug) screen (UDS) must be negative for any substance for which the subject does not have a valid prescription.

#### Medical Criteria

- 6. Has developed a serious and/or unstable psychiatric, neurologic, cardiovascular (e.g., long QT syndrome, torsade de pointes, unstable cardiac syndrome or syncope, congestive heart failure, ongoing uncorrected hypokalemia or hypomagnesemia, non-sustained or sustained ventricular tachycardia), respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies that, in the judgment of the Investigator, would jeopardize the safe participation of the subject in the study, or has major surgery planned during the study
- 7. Has experienced any change in medical or treatment status that may increase the risk associated with taking pimavanserin, would interfere with safety assessments, or would confound the interpretation of study results, based on the Investigator's judgment
- 8. For age <13 years, a resting position (sitting or supine) systolic (SBP) and/or diastolic blood pressure (DBP) level ≥90th percentile for gender-specific age and height charts from the National Heart and Lung Institute (NHLI), at Baseline. For age ≥13 years a resting position (sitting or supine) SBP ≥120 mmHg and/or a DBP ≥80 mmHg, at Baseline.
- 9. Has a clinically significant abnormal ECG at Baseline or any of the following cardiac conduction abnormalities:
  - a. Corrected QT interval using Fridericia's correction method (QTcF) ≥450 ms
  - b. PR interval on ECG >220 ms

| | c. Evidence of second- or third-degree atrioventricular block |
|---|---|
| | d. Evidence of complete left bundle branch block |
| | e. Intraventricular conduction delay with QRS interval on ECG (QRS) >110 ms |
| | f. QRS or T wave morphology that could, in the Investigator's opinion, render QT interval assessment unreliable |
| | g. Sick sinus syndrome |
| | h. Non-sinus rhythm |
| | i. Resting heart rate <50 beats per minute |
| | One repeat set of triplicate ECGs is allowed at Baseline. |
| | 10. Weight <15 kg |
| | 11. <i>In Italy only</i> : Has a sensitivity to any compound present in pimavanserin or any metabolites or compounds listed in the Investigator's brochure as being present in this medication |
| Sample size calculations | The planned sample size for this study is not based on statistical power but will depend on the number of subjects who complete the antecedent double-blind study, and who rollover into this open-label extension study. |
| Statistical methods | The primary objective of this study is to evaluate the long-term safety and tolerability of pimavanserin after 52 weeks of treatment in children and adolescents with ASD. Secondary and exploratory objectives include assessment of efficacy outcome measures over time. No formal statistical testing will be performed for any of the safety or efficacy endpoints. |
| | All safety and efficacy measures will be summarized using descriptive statistics. |
| | For each continuous measure in safety and efficacy analyses, changes from Baseline results will be presented in two ways: |
| | using the Baseline of this study to report the changes across the timepoints of this open-label study |

2. using the Baseline from the antecedent doubleblind study to report the changes across the timepoints of this open-label study


Date: 29 February 2024

## **Descriptive Statistics**

For continuous variables, the following summary statistics will be provided: number of subjects, mean, standard error of the mean, standard deviation, minimum, maximum, and median. For categorical variables, summaries will include the number and percentage of subjects in each category.

## **Population Analysis Sets**

The **Safety Analysis Set** will include all subjects who received at least one dose of open-label study drug. The Safety Analysis Set will be used for all analyses.

#### Subgroup Analysis

Selected analyses may be performed in subgroups defined in the statistical analysis plan (SAP).

#### **Missing Data**

Handling of missing values will be described in detail in the SAP.

#### **Primary Analyses**

The primary endpoints for this study are TEAEs. All adverse events will be classified into standard terminology using the Medical Dictionary for Regulatory Activities (MedDRA). The number and frequency of TEAEs will be summarized by system organ class and preferred term. TEAEs leading to discontinuation, TEAEs related to study drug, TEAEs by maximum severity, fatal TEAEs, serious TEAEs, and serious TEAEs related to study drug will also be summarized.

#### **Other Safety Analyses**

Descriptive statistics for ECGs, vital signs, weight, BMI, ESRS-A, and clinical laboratory parameters, including changes from Baseline, will be tabulated by timepoint. Additionally, categorical analyses will be conducted on the incidence of subjects with prolonged corrected QT interval on ECG (QTc) intervals and changes in QTc intervals in accordance with International Council for Harmonisation (ICH) guidelines.

| | For the C-SSRS, the number and percentage of subjects with suicidal ideation or behavior during the study will be tabulated. |
|---|---|
| | Efficacy Analyses |
| | Descriptive statistics for all efficacy endpoints will be tabulated by timepoint. |
| Date | 29 February 2024 |





Abbreviations: EOT=end of treatment; ET=early termination; yrs=years

<sup>&</sup>lt;sup>a</sup> A dose increase, based on the Investigator's assessment of clinical response, may be made at the Week 2 visit. After the Week 2 visit and up to and including the Week 20 visit, dose adjustments, either increases or decreases, may be made at any clinic visit (scheduled or unscheduled), based on the Investigator's assessment of clinical response and tolerability. No further dose adjustments are allowed after the Week 20 visit.

Table S-1 Schedule of Events and Assessments for ACP-103-070

| Period | | Open-label treatment period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline <sup>w</sup> | | | | | | | | EOT/ET <sup>n</sup> | Unscheduled <sup>a</sup> | Safety<br>follow-up <sup>b</sup> |
| Visit Week | 0 | 2 | 6 | 12 | 20 | 28 | 36 | 44 | 52 | | 56 |
| Visit number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | 10 |
| Visit window (days) | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | | +3 |
| Type of visit <sup>c</sup> | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Telephone |
| Informed consent/assent <sup>d</sup> | X | | | | | | | | | | |
| Inclusion/exclusion criteria | Xe | | | | | | | | | | |
| Physical examination and self- or caregiver-reported Tanner staging <sup>q</sup> | X | | | X | | X | | X | X | | |
| Vital signs | X | X | X | X | X | X | X | X | X | X | |
| Height <sup>s</sup> , weight, and BMI | X | X | X | X | X | X | X | X | X | X | |
| 12-lead ECG <sup>f, g, m</sup> | X | X | X | X | X | X | X | X | X | | |
| Clinical laboratory tests <sup>g, m, r, v, x</sup> | X | | | X | | X | | X | X | | |
| Pregnancy test <sup>g, h</sup> | X | X | X | X | X | X | X | X | X | X | |
| Urine toxicology (drug) screen (UDS)° | X | | | | | | | | X | | |
| ABCq | X | X | X | X | X | X | X | X | X | | |
| CGI-S of irritability | X | X | X | X | X | X | X | X | X | | |
| CGI-I of irritability <sup>i</sup> | X | X | X | X | X | X | X | X | X | | |
| RBS-R <sup>q</sup> | X | | | X | | X | X | X | X | | |
| VABS-Socialization <sup>q</sup> | X | | | X | | X | X | X | X | | |

Table continues on next page

Table S-1 Schedule of Events and Assessments for ACP-103-070 (Continued)

| Period | | Open-label treatment period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baselinew | | | | | | | | EOT/ET <sup>n</sup> | Unscheduled <sup>a</sup> | Safety<br>follow-up <sup>b</sup> |
| Visit Week | 0 | 2 | 6 | 12 | 20 | 28 | 36 | 44 | 52 | | 56 |
| Visit number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | 10 |
| Visit window (days) | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | | +3 |
| Type of visit <sup>c</sup> | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Clinic | Telephone |
| CGSQ <sup>q</sup> | X | | X | | X | X | X | X | X | | |
| C-SSRS <sup>q</sup> | X | X | X | X | X | X | X | X | X | X | |
| ESRS-A <sup>q</sup> | X | X | X | X | X | X | X | X | X | X | |
| Assessment of concomitant medications <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Assessment of adverse events | X | X | X | X | X | X | X | X | X | X | X |
| Assessment of syncope occurrence <sup>t</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Assessment of somnolence occurrence <sup>u</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Study drug dispensation | $X^{j}$ | X | X | X | X | X | X | X | | $X^k$ | |
| Study drug return and accountability <sup>1</sup> | | X | X | X | X | X | X | X | X | X | |

Abbreviations: ABC=Aberrant Behavior Checklist; ASR=accurate symptom reporting; BMI=body mass index; CGI-I=Clinical Global Impression–Improvement; CGI-S=Clinical Global Impression–Severity; CGSQ=Caregiver Strain Questionnaire; C-SSRS=Columbia–Suicide Severity Rating Scale; ECG=electrocardiogram; eGFR=estimated glomerular filtration rate; EOT=end of treatment; ESRS-A=Extrapyramidal Symptom Rating Scale–Abbreviated; ET=early termination; LAR=legally acceptable representative; RBS-R= Repetitive Behavior Scale–Revised; UDS=urine toxicology (drug) screen; VABS=Vineland Adaptive Behavior Scales

- At a minimum the safety assessments indicated should be completed at unscheduled visits. Other assessments may be completed at unscheduled visits at the discretion of the Investigator.
- This visit is a safety follow-up telephone call visit for subjects who complete the study or discontinue treatment prematurely from the study. This visit will occur 30(+3) days after the last dose of study drug. The safety follow-up visit will not be done if the subject withdraws consent to participate in all parts of the study.
- <sup>c</sup> Circumstances may arise (e.g., pandemic, natural disaster, political upheaval, or to minimize subject and caregiver burden) when on-site assessments of efficacy and/or safety are not possible. In those cases, assessments may be performed offsite by raters either in person, or via video technology or telephone

where possible. For all visits that are conducted remotely, the Investigator <u>must</u> contact the Medical Monitor for approval of the plan. Sites must keep a log to identify details of all visits that are administered remotely. Provided that the subject is physically in the clinic, and accompanied by a relative, all caregiver-rated assessments may be provided remotely.

- d Consent from the subject, parent/LAR, and caregiver (if different from the parent/LAR), for the present study must be obtained for entry into the present study prior to the final procedures being performed at the end of treatment (EOT) visit in the antecedent double-blind study. Data from the EOT/ET visit procedures of the antecedent double-blind study will be carried over as baseline information in the present study, as applicable
- <sup>c</sup> All assessments must be completed and subject must meet required eligibility criteria before being enrolled.
- 12-lead ECGs should be performed in sequential triplicate. Electrocardiograms should be performed before blood sampling or at least 30 minutes after blood sampling. The subject must rest in a sitting or supine position for 5 minutes before the ECG is obtained. One repeat set of triplicate ECGs is allowed at Baseline.
- Mild sedation is allowed exceptionally for ECGs and blood draws during the study (e.g., alprazolam at a pediatric-appropriate dose per age, and the *lowest dose* deemed necessary by the Investigator) just in cases when the subject's agitation/anxiety does not allow a safe and accurate measurement and the Investigator, with agreement from the caregiver, considers it safe and appropriate for the subject.
- For female subjects of childbearing potential, a urine pregnancy dipstick test will be completed at all scheduled and unscheduled visits. If positive, the result will be confirmed with a serum pregnancy test.
- Relative to baseline status in the antecedent double-blind study.
- The subject and their parent/LAR will be provided instructions for the subject's first dose of study drug on the day after the Baseline visit.
- k Study drug may be dispensed to the subject at unscheduled visits if needed.
- If visit is remote, accountability will be assessed verbally with the caregiver, and verified at the next clinic visit.
- The involvement of experienced personnel in the conduction of routine procedures such as blood drawing and ECG recording in this population is strongly recommended.
- The ET visit will not be done if the subject (and/or parent/LAR) withdraws consent to participate in all parts of the study and withdrawal of consent happens before that timepoint.
- <sup>o</sup> A urine toxicology dipstick should be used in addition to the urine toxicology screen at the Baseline visit (to confirm eligibility).
- p Including coronavirus disease 2019 (COVID-19) vaccination
- For scales that require caregiver input, the caregiver should be the parent/LAR or designee. A designee should be a family member, adult and responsible, living with or in very frequent contact with the subject participating in the study, who is committed to providing responses for the caregiver-reported scales for the duration of Studies ACP-103-069 and ACP-103-070. Caregivers providing input for the ABC, RBS-R, and CGSQ scales will be trained in accurate symptom reporting (ASR) prior to completing the scales. ASR training should be done at Screening in the antecedent study (Study ACP-103-069) before the caregiver completes any scales, and repeated whenever there is a change in caregiver or if the site feels a caregiver requires retraining.
- Prolactin CCI Results will be monitored CCI
- s As measured by stadiometer.
- If the caregiver reports an occurrence of syncope, the investigator should ask the "syncope adverse event questions" in Appendix G.
- <sup>u</sup> If the caregiver reports an occurrence of somnolence, the investigator should ask the "somnolence adverse event questions" in Appendix H.


Study: ACP-103-070 Final Version: 2.0 Date: 29 February 2024

- Circumstances may arise (e.g., pandemic, natural disaster, political upheaval, or technical issues) when on-site clinical laboratory tests are not possible. In those cases, clinical laboratory tests may be performed at the subject's place of residence by study staff or at a local laboratory. The Investigator must contact the Medical Monitor for approval with the plan. Sites must keep a log to identify details of all visits that are administered remotely.
- Procedures performed at the EOT visit for Study ACP-103-069 will be carried over as baseline information, if applicable.
- In Italy only: CCI

# TABLE OF CONTENTS

| SPONSO | R SIGNATURE PAGE | 2 |
|---|---|---|
| DECLAR | ATION OF INVESTIGATOR | 4 |
| PROTOC | COL SYNOPSIS | 5 |
| TABLE C | OF CONTENTS | 21 |
| LIST OF | TABLES | 26 |
| LIST OF | FIGURES | 26 |
| LIST OF | ABBREVIATIONS AND DEFINITION OF TERMS | 27 |
| 1 | INTRODUCTION | 29 |
| 1.1 | Background Information | 29 |
| 1.1.1 | Autism Spectrum Disorder | 29 |
| 1.1.2 | Current Treatments for Irritability Associated With Autism Spectrum Disorder | 29 |
| 1.1.3 | Scientific Rationale | |
| 1.2 | Investigational Product | 32 |
| 1.3 | Previous Clinical Experience | 32 |
| 1.3.1 | Studies in Adults With Schizophrenia | 33 |
| 1.3.2 | Phase 1 Study in Adolescents With Psychiatric Disorders | |
| 1.4 | Study Rationale | 35 |
| 1.4.1 | Rationale for Study Design | |
| 1.4.2 | Rationale for Dose Selection | |
| 1.5 | Benefit/Risk Assessment | |
| 1.5.1 | Known Potential Risks | |
| 1.5.2 | Known Potential Benefits. | |
| 2 | STUDY OBJECTIVES AND ENDPOINTS | |
| 2.1 | Primary Objective. | |
| 2.1.1 | Primary Endpoints | |
| 2.2 | Secondary Objective | |
| 2.2.1 | Secondary Endpoint | |
| 2.3 | Exploratory Objectives | |
| 2.3.1 | Exploratory Endpoints. | |
| 3 | STUDY DESCRIPTION | |
| 3.1 | Overview of Study Design | |
| 3.1.1 | Open-label Treatment Period (52 Weeks) | |
| 3.1.2 | Safety Follow-up Period (30 Days) | 41 |


| 4 | SUBJECT ELIGIBILITY AND WITHDRAWAL CRITERIA | 41 |
|---|---|---|
| 4.1 | Inclusion Criteria | 42 |
| 4.2 | Exclusion Criteria | 43 |
| 4.3 | Screen Failures | 45 |
| 4.4 | Subject Withdrawal of Consent | 45 |
| 4.5 | Subject Discontinuation | 45 |
| 4.5.1 | Handling of Subject Discontinuation During the Treatment Period | |
| 4.6 | Subject Lost to Follow-up | |
| 4.7 | Study Discontinuation | 46 |
| 4.8 | Prior and Concomitant Therapy | 47 |
| 4.8.1 | Prior Medication | |
| 4.8.2 | Concomitant Medication | |
| 4.8.2.1 | Permitted, Restricted, and Prohibited Medications | 47 |
| 4.8.3 | Rescue Medications, Treatments, and Procedures | 48 |
| 5 | INVESTIGATIONAL PRODUCT | 48 |
| 5.1 | Investigational Product Description | 48 |
| 5.1.1 | Formulation, Appearance, Packaging, and Labeling | 48 |
| 5.1.2 | Product Storage and Stability | |
| 5.1.3 | Dosing and Administration | 49 |
| 5.1.3.1 | Dose Modification | 49 |
| 5.1.4 | Blinding | 49 |
| 5.1.5 | Study Drug Compliance | 49 |
| 5.1.6 | Overdose | 50 |
| 5.2 | Investigational Product Accountability Procedures | 50 |
| 6 | STUDY ASSESSMENTS | 50 |
| 6.1 | Baseline Assessments | 51 |
| 6.1.1 | Physical Examination and Self- or Caregiver-reported Tanner Staging | 51 |
| 6.1.2 | Vital Signs | 51 |
| 6.1.3 | Height, Weight, and Body Mass Index | 51 |
| 6.1.4 | 12-lead ECG | 51 |
| 6.1.5 | Clinical Laboratory Tests | 51 |
| 6.1.6 | Pregnancy Test | 51 |
| 6.1.7 | Urine Toxicology (Drug) Screen | 51 |
| 6.1.8 | Aberrant Behavior Checklist | 51 |
| 6.1.9 | CGI-S | 52 |
| 6.1.10 | CGI-I | 52 |

| 6.1.11 | RBS-R | 52 |
|---|---|---|
| 6.1.12 | VABS-Socialization | 52 |
| 6.1.13 | CGSQ | 52 |
| 6.1.14 | C-SSRS | 52 |
| 6.1.15 | ESRS-A | 52 |
| 6.1.16 | Concomitant Medications and Adverse Events | 52 |
| 6.2 | Efficacy Assessments | 52 |
| 6.2.1 | Aberrant Behavior Checklist | 52 |
| 6.2.2 | CGI-S | 53 |
| 6.2.3 | CGI-I | 53 |
| 6.2.4 | Repetitive Behavior Scale–Revised | 53 |
| 6.2.5 | Vineland Adaptive Behavior Scales–Socialization | |
| 6.2.6 | Caregiver Strain Questionnaire | |
| 6.3 | Safety Scales | 55 |
| 6.3.1 | Columbia-Suicide Severity Rating Scale. | 55 |
| 6.3.2 | Extrapyramidal Symptom Rating Scale-Abbreviated | |
| 6.4 | Safety Assessments | 56 |
| 6.4.1 | Physical Examination and Self- or Caregiver-reported Tanner Staging | 56 |
| 6.4.2 | Vital Signs | 57 |
| 6.4.3 | Electrocardiograms | 57 |
| 6.4.4 | Laboratory Evaluations | 58 |
| 6.4.5 | Syncope | 60 |
| 6.4.6 | Somnolence | 60 |
| 6.5 | Blood Sampling | 61 |
| 6.6 | Safety Follow-up | 62 |
| 6.7 | Unscheduled Visits | 63 |
| 6.8 | Remote Assessments or Visits | 63 |
| 7 | ADVERSE EVENTS | 63 |
| 7.1 | Specification of Safety Parameters | 63 |
| 7.1.1 | Definition of Adverse Event | 63 |
| 7.1.2 | Definition of Serious Adverse Event | 64 |
| 7.2 | Classification of an Adverse Event | 65 |
| 7.2.1 | Severity of Event | 65 |
| 7.2.2 | Relationship to Study Drug | 65 |
| 7.2.3 | Duration | 66 |
| 7.2.4 | Frequency | 66 |

| 7.2.5 | Action Taken With Study Drug | 66 |
|---------|--------------------------------------------------------------|----|
| 7.2.6 | Therapy | 67 |
| 7.2.7 | Outcome | 67 |
| 7.2.8 | Seriousness | 67 |
| 7.2.9 | Definition of Unexpectedness | 67 |
| 7.3 | Time Period and Frequency for Event Assessment and Follow-up | 67 |
| 7.4 | Reporting Procedures | 67 |
| 7.4.1 | Adverse Event Reporting | 67 |
| 7.4.2 | Serious Adverse Event Reporting | 68 |
| 7.4.3 | Reporting of Pregnancy | 69 |
| 7.4.3.1 | Reporting Paternal Drug Exposure | 69 |
| 7.4.4 | Reporting of Overdose | 69 |
| 8 | MONITORING | 69 |
| 9 | STATISTICAL METHODS AND DATA ANALYSIS | 70 |
| 9.1 | Statistical and Analytical Plans | 70 |
| 9.2 | Statistical Hypotheses | 70 |
| 9.3 | Sample Size Determination | 70 |
| 9.4 | Population Analysis Sets | 70 |
| 9.5 | Statistical Analyses | 70 |
| 9.5.1 | Primary Analyses | 71 |
| 9.5.2 | Other Safety Analyses | 71 |
| 9.5.3 | Secondary Endpoint and Analysis | 71 |
| 9.5.4 | Exploratory Endpoints and Analyses | 71 |
| 9.5.5 | Subgroup Analyses | 72 |
| 9.6 | Interim Analyses | 72 |
| 9.7 | Data and Safety Monitoring Board | 72 |
| 10 | STUDY MANAGEMENT AND DATA COLLECTION | 72 |
| 10.1 | Data Collection and Management Responsibilities | 72 |
| 10.2 | Source Documents | 73 |
| 10.3 | Case Report Forms | 73 |
| 10.4 | Confidentiality | 73 |
| 10.5 | Study Records Retention | 73 |
| 10.6 | Protocol Exceptions and Deviations | 74 |
| 10.7 | Protocol Amendments | 74 |
| 11 | QUALITY MANAGEMENT | 74 |

| 11.1 | Risk Management | ļ |
|---|---|---|
| 11.2 | Quality Control and Quality Assurance | 5 |
| 12 | ETHICAL CONSIDERATIONS | 5 |
| 12.1 | Ethical Standard | 5 |
| 12.2 | Institutional Review Board/Ethics Committee | 5 |
| 12.3 | Informed Consent/Assent Process | 5 |
| 12.3.1 | Subject Assent Form | 7 |
| 12.3.2 | Parent and Legally Acceptable Representative Informed Consent | 7 |
| 12.3.3 | Consent and Other Informational Documents Provided to Subjects | 7 |
| 12.3.4 | Consent Procedures and Documentation | 7 |
| 12.3.4.1 | Remote Consent Procedures and Documentation | 3 |
| 13 | PUBLICATION PLAN | 3 |
| 14 | CONFLICT OF INTEREST POLICY | 3 |
| 14.1 | Finance, Insurance, and Indemnity | 3 |
| 15 | LITERATURE REFERENCES | ) |
| 16 | APPENDICES83 | Ĺ |
| Appendix | A Prohibited and Restricted Medications <sup>a</sup> | Ĺ |
| Appendix | B Prohibited and Restricted Concomitant Medications: Inhibitors and Inducers of Cytochrome P450 Enzyme 3A4 | 5 |
| Appendix | C Criteria for Identifying Potentially Clinically Important Laboratory Values88 | 3 |
| Appendix | D Criteria for Potentially Clinically Important ECG Values | ) |
| Appendix | E Criteria for Identifying Additional ECG Measurements of Potential Clinical Relevance. To be Used for Medical Monitoring Purposes90 | ) |
| Appendix | F Criteria for Potentially Clinically Important Vital Signs | Ĺ |
| Appendix | G Syncope Adverse Event Questions | 2 |
| Appendix | H Somnolence Adverse Event Questions | 3 |

# LIST OF TABLES

| Table S-1 | Schedule of Events and Assessments for ACP-103-070 | 17 |
|---|---|---|
| Table 6–1 | Safety Laboratory Evaluations | 60 |
| Table 6–2 | Blood Collection Volume Limits in Affected Children | 61 |
| Table 6–3 | Blood Collection Volumes for Safety Labs (6- through 17-year-olds) | 62 |
| Table 6–4 | Blood Collection Volumes for Safety Labs (5-year-olds) | 62 |
| | LIST OF FIGURES | |
| Figure S–1 | Schematic of Study Design for ACP-103-070 | 16 |

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Term | Definition |
|---|---|
| 5-HT | 5-hydroxytryptamine (serotonin) |
| 5-HT <sub>2A</sub> receptor | 5-hydroxytryptamine (serotonin) receptor subtype 2A |
| 5-HT <sub>2C</sub> receptor | 5-hydroxytryptamine (serotonin) receptor subtype 2C |
| ABC | Aberrant Behavior Checklist |
| ABC-I | Aberrant Behavior Checklist–Irritability |
| AC-279 | N-desmethyl-pimavanserin, major metabolite of pimavanserin |
| AE | adverse event |
| ASD | autism spectrum disorder |
| ASR | accurate symptom reporting |
| AUC | area under the plasma concentration-time curve |
| $\mathrm{AUC}_{	au}$ | area under the plasma concentration-time curve during any dosing interval at steady state |
| BMI | body mass index |
| CGI-I | Clinical Global Impression-Improvement |
| CGI-S | Clinical Global Impression-Severity |
| CGSQ | Caregiver Strain Questionnaire |
| CFR | Code of Federal Regulations |
| C <sub>max</sub> | maximum (peak) observed drug concentration |
| C <sub>max-ss</sub> | C <sub>max</sub> at steady state |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| DSMB | data and safety monitoring board |
| EC | ethics committee |
| ECG | Electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| eGFR | estimated glomerular filtration rate |
| EOT | end of treatment |
| ESRS-A | Extrapyramidal Symptom Rating Scale–Abbreviated |
| ET | early termination |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HDL | high-density lipoprotein |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IRB | institutional review board |


| Term | Definition |
|--------|------------------------------------------------------------|
| LAR | legally acceptable representative |
| NSA-16 | Negative Symptom Assessment–16 |
| PANSS | Positive and Negative Syndrome Scale |
| PDP | Parkinson's disease psychosis |
| PK | pharmacokinetic(s) |
| QD | once daily |
| QRS | QRS interval on ECG |
| QT | QT interval on ECG |
| QTc | corrected QT interval on ECG |
| QTcF | corrected QT interval using Fridericia's correction method |
| RBS-R | Repetitive Behavior Scale–Revised |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| TEAE | treatment-emergent adverse event |
| US | United States |
| VABS | Vineland Adaptive Behavior Scales |

#### 1 INTRODUCTION

This document is a research protocol and the described study will be conducted in compliance with the protocol, the International Council for Harmonisation (ICH) Good Clinical Practice (GCP) Guideline, and applicable regulatory requirements.

## 1.1 Background Information

### 1.1.1 Autism Spectrum Disorder

Autism spectrum disorder (ASD) is a heterogeneous neurodevelopmental disorder characterized by impairments in social interactions, communication, and restricted interests and stereotyped behaviors. In 2014, the Centers for Disease Control and Prevention (CDC) estimated that an average of 1 in 59 children in the United States (US) has an ASD. In the Diagnostic and Statistical Manual of Mental Disorders—Fifth Edition (DSM-5) criteria, ASD includes autistic disorder, Asperger's syndrome, pervasive developmental disorder-not otherwise specified (PDD-NOS), and childhood disintegrative disorder (Grzadzinski et al. 2013). The etiology of ASD is highly genetic although environmental factors also contribute. Heritability estimates from family and twin studies suggest that about 90% of variance can be attributed to genetic factors, making ASD the neuropsychiatric disorder most affected by genetic factors (Levy et al. 2009). Core symptoms of ASD are usually observed by 3 years of age, although typical language development might delay the diagnosis of ASD.

Beyond the variability in the presentation of core symptoms of ASD, affected individuals also vary with respect to associated non-ASD symptoms. Both cognitive and intellectual disabilities often coexist with language deficits, motor abnormalities, attentional difficulties, hyperactivity, and sleep disruptions. Seventy-five percent of ASD patients suffer from comorbid psychiatric conditions, but also a number of medical comorbidities. While the association between comorbidities and the severity of autism-related symptoms remains unclear (Aldinger et al. 2015), the clinical picture of severe irritability and behavioral problems, aggravated by the child's inability to verbally express discomfort or anxiety, causes families and peers greater distress and requires treatment.

#### 1.1.2 Current Treatments for Irritability Associated With Autism Spectrum Disorder

At present, no pharmacological treatment has been Food and Drug Administration (FDA) approved for treatment of core deficits in ASD. Both pharmacological and nonpharmacological interventions that provide partial symptomatic relief of core and associated symptoms are seen in clinical practice. Pharmacological treatments include psychostimulants, atypical antipsychotics, antidepressants, and alpha-2 adrenergic receptor agonists (Sharma et al. 2018). In the absence of methods to identify specific behavioral phenotypes with shared underlying pathophysiology to develop targeted treatment, management of irritability and maladaptive, self-injurious behaviors


regardless of their underlying cause becomes a priority. Consequently, the only two FDA approved drugs, indicated for treatment of irritability associated with autistic disorder in children and adolescents 5 to 17 years of age (6 to 17 years for aripiprazole, 5 to 16 years for risperidone), are Risperdal® (risperidone) and Abilify® (aripiprazole). However, both are associated with a number of serious side effects of which significant weight gain and metabolic side-effects are particularly prominent (McPheeters et al. 2011). Accordingly, there is a high unmet medical need for pharmacological treatments of both core and associated symptoms of the disorder that would have better efficacy and safety and tolerability profile.

#### 1.1.3 Scientific Rationale

Pimavanserin exerts its antipsychotic activity as an inverse agonist/antagonist (Vanover et al. 2006) at 5-hydroxytryptamine (serotonin) receptor subtype 2A (5-HT<sub>2A</sub>) receptors, and to a lesser extent at 5-hydroxytryptamine (serotonin) receptor subtype 2C (5-HT<sub>2C</sub>) receptors. Both risperidone and aripiprazole are dopamine type-2 (D<sub>2</sub>) receptor antagonists but also have 5-HT<sub>2A</sub> receptor antagonist activity (risperidone is also an inverse 5-HT<sub>2A</sub> agonist) and are approved for the treatment of irritability and behavioral symptoms in children with autism. Irritability associated with ASD is often caused by multiple underlying comorbid conditions (anxiety, sleep disorders, mood instability due to epilepsy, etc.) many of which are linked to serotonergic system dysfunction).

The serotonin system has long been implicated in autism spectrum disorder by both peripheral and brain findings (Muller et al. 2016). In people with autism, brain activation differences of inhibitory control regions are differentially modulated by serotonin, and may partially underpin some of the core and associated symptoms of ASD (Daly et al. 2014). Consequently, while the underlying mechanism of irritability is not well established, it is possible that such modulation of the serotonergic system, a property shared by pimavanserin and two approved antipsychotics, is associated with the treatment effect on irritability associated with ASD. The involvement of neurotransmitters such as 5-hydroxytryptamine (serotonin) (5-HT) has been suggested previously in autistic disorder as increased platelet 5-HT levels were found in 40% of the autistic population, suggesting that hyperserotonemia may be a pathologic factor in infantile autism. Alterations in platelet serotonin 5-HT<sub>2A</sub> binding were also detected (Aaron et al. 2019). Perhaps one of the earliest neurochemical investigations of autism suggested that the mean level of 5-HT in the whole blood of autistic children was elevated compared to levels in non-autistic children (Ritvo et al. 1970; Rolf et al. 1993). The many repeated observations of this difference have led to the "hyperserotonin hypothesis of autism" hypothesizing that ASD behavior is a consequence of some defect in tryptophan or 5-HT biochemistry in specific brain regions. Both ritanserin and cyproheptadine, two known 5-HT<sub>2</sub> receptor antagonists, have been tried as monotherapy and adjunct therapy in children with irritability associated with ASD. A positive


2004).

effect of ritanserin, a selective 5-HT<sub>2</sub> receptor antagonist, in children with ASD and mental retardation was reported mostly in reduction of psychomotor instability and impaired concentration and attention (Paclt and Hellerová 1993). Likewise, improvement in disruptive behavior was seen in an adjunctive treatment study with cyproheptadine (Akhondzadeh et al.

Studies in rodent models also demonstrate that the serotonin system is involved in both social function and repetitive behavior, the two core symptom domains of ASD. Importantly, risperidone and aripiprazole, both of which have significant action on the serotonin 5-HT<sub>2A</sub> receptor as inverse agonists/antagonists, have shown improvement in repetitive behaviors as a side benefit when used to treat irritability/agitation (Fung et al. 2016).

Hence, considering that pimavanserin is a more selective 5-HT<sub>2A</sub> inverse agonist/antagonist without measurable activity at dopaminergic, histaminergic, adrenergic, or muscarinic receptors, it is plausible that pimavanserin would show efficacy (and potentially better tolerability due to reduced off-target effects) in the treatment of irritability associated with ASD. This is particularly important as children with autism usually have medical comorbidities and may be more sensitive to the side effects of medications especially in the context of polypharmacy. Beneficial effects on some of the core symptoms of ASD may also be anticipated given its 5-HT<sub>2A</sub> activity.

#### **Supportive Pimavanserin Data**

Although the data from recently completed adult adjunctive studies in schizophrenia provide limited evidence of efficacy on symptoms of interest in ASD, directly selective 5-HT<sub>2A</sub> inverse agonists like pimavanserin improve slow wave sleep, restore circadian rhythms, and may thereby alleviate irritability. It is proposed that pimavanserin's downregulation of 5-HT<sub>2A</sub>-induced anxiety, supported by data from Study ACP-103-042 in patients with major depressive disorder and an inadequate response to antidepressant therapy, may improve depression and anxiety often present with a clinical picture of irritability in the pediatric population with ASD. The potential efficacy in social deficits has been demonstrated in greater efficacy in the social involvement domain of the Negative Symptom Assessment–16 (NSA-16) in the recently completed study adjunctive treatment of negative symptoms of schizophrenia. Finally, pimavanserin does not exert troublesome and persistent sedative effects that would impact overall functioning or already challenging school performance in this population.

Pimavanserin's lack of off-target activity that supports its use in this vulnerable pediatric population. Both short- and long-term data from completed adult studies with pimavanserin as monotherapy and in an adjunctive setting confirm its benign safety profile and consistent side effect profile. In comparison to the other approved antipsychotics, there has been no or negligible impact on weight, metabolic parameters, or extrapyramidal changes, and the impact on corrected


Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

QT interval on ECG (QTc) prolongation even with the maximum pimavanserin dose has been minimal.

#### 1.2 **Investigational Product**

Pimavanserin is an atypical antipsychotic that is present in the investigational product (IP) as pimavanserin tartrate salt with the chemical name, urea, N-[(4-fluorophenyl)methyl]-N-(1methyl-4-piperidinyl)-N'-[[4-(2-methylpropoxy)phenyl]methyl]-, (2R,3R)-2,3dihydroxybutanedioate (2:1). In April 2016, pimavanserin was approved in the US for the treatment of hallucinations and delusions associated with Parkinson's disease psychosis (PDP).

Pimavanserin is a novel small molecule designed to specifically block serotoninergic neurotransmission mediated by the 5-HT<sub>2A</sub> receptor. At higher doses, pimavanserin may block 5-HT<sub>2C</sub> receptors (Vanover et al. 2006). Pimavanserin shows no appreciable activity at dopaminergic, adrenergic, histaminergic, or muscarinic receptors in vitro. On the basis of its novel receptor binding profile, pimavanserin may have benefits with regard to overall tolerability relative to other antipsychotic agents.

#### 1.3 **Previous Clinical Experience**

Always refer to the latest version of the pimavanserin Investigator's Brochure for the overall benefit/risk assessment and the most accurate and current information regarding non-clinical data, drug metabolism, pharmacokinetics (PK), efficacy, and safety.

The clinical PK, pharmacodynamics, efficacy, and safety of pimavanserin have been evaluated in a total of 34 completed studies, four studies in reporting, nine otherwise ongoing studies, and one completed expanded-access program (EAP). As of 28 April 2020, approximately 3594 subjects had been exposed to pimavanserin, including 552 healthy subjects, 12 renally impaired subjects, 25 hepatically impaired subjects, 34 adolescents with psychiatric disorders, 711 subjects with Parkinson's disease/PDP (of which 632 had PDP, including 15 in the EAP), 90 subjects with Alzheimer's disease psychosis, 96 subjects with agitation and aggression in Alzheimer's disease, 392 subjects with dementia-related psychosis, 433 subjects in additional studies in frail subjects with neurodegenerative disease and neuropsychiatric symptoms, 909 subjects diagnosed with schizophrenia, and 340 subjects with major depressive disorder.

According to the most recent estimate (28 April 2020), at least 32,291 patients have received NUPLAZID® (pimavanserin) commercially, representing 21,001 person-years of exposure.

Pimavanserin is considered to be generally safe and well tolerated. In single and multiple dose studies in healthy subjects, the highest doses administered were 255 mg and 136 mg/day, respectively.

Clinical Study Protocol Amendment 3-Consolidated

#### 1.3.1 Studies in Adults With Schizophrenia

The use of pimavanserin in schizophrenia has been evaluated in three Phase 2 studies (ACP-103-007, ACP-103-008, and ACP-103-038) and one Phase 3 study (ACP-103-034). Patients completing ACP-103-034 and ACP-103-038 also had the opportunity to enroll in an ongoing open-label extension study (ACP-103-035).

Studies ACP-103-007 and ACP-103-008 evaluated the efficacy of pimavanserin as concomitant therapy (with risperidone or haloperidol) in subjects with schizophrenia. Results of Study ACP-103-007 suggested a rapid onset of anti-akathisia effects with pimavanserin treatment (difference from placebo not statistically significant), without affecting haloperidol concentrations. Study ACP-103-008 demonstrated that pimavanserin 17 mg plus 2 mg risperidone was significantly more efficacious than 2 mg risperidone plus placebo and similar in efficacy to standard (6 mg) risperidone. Pimavanserin 17 mg plus 2 mg risperidone appeared to demonstrate greater efficacy at Day 15 than either 2 mg risperidone plus placebo or 6 mg risperidone plus placebo (or 2 mg haloperidol plus placebo).

Study ACP-103-034 was a Phase 3, 6-week, randomized, double-blind, placebo-controlled study in outpatients with schizophrenia with an inadequate response to current antipsychotic treatment. A total of 396 subjects (198 per treatment group) were randomized across 88 sites in Europe and North America. Subjects were randomized to receive up to 6 weeks of adjunctive placebo or pimavanserin, at 20 mg once daily (QD) for Week 1, remaining at 20 mg or adjusted to 10 or 34 mg QD over the next 2 weeks, and remaining at the same dose for the last 3 weeks. Of the 396 randomized subjects, 364 (91.9%) completed the study, including 190 (96.0%) in the placebo group and 174 (87.9%) in the pimavanserin group.

Adding pimavanserin to existing antipsychotic treatment resulted in improvement of psychotic symptoms. The change from Baseline to Week 6 on the primary efficacy endpoint (Positive and Negative Syndrome Scale [PANSS] total score) was numerically greater in the pimavanserin group (-15.3) than in the placebo group (-13.4), although the difference was not statistically significant (mixed-effect model repeated measures [MMRM] least squares mean [LSM] difference: -2.1, 95% CI -4.5, 0.4, p=0.0940; Cohen's d=0.173). A positive trend was observed on the key secondary endpoint, the change from Baseline to Week 6 in Clinical Global Impression-Severity (CGI-S) score.

In the prespecified subgroup analysis by region, consistent positive results were observed for subjects enrolled in Europe on both the primary endpoint, PANSS total score (unadjusted p=0.0234), and the key secondary endpoint, CGI-S score (unadjusted p=0.0214).

Notable improvements in favor of pimavanserin were seen on prespecified measures of negative symptoms: the secondary endpoint PANSS negative subscale score (unadjusted p=0.0474) and


the exploratory endpoint PANSS Marder Negative Symptoms Factor score (unadjusted p=0.0362). Numerical difference in favor of pimavanserin was also seen in the change from Baseline to Week 6 in Karolinska Sleepiness Scale score (unadjusted p=0.0265).

Study ACP-103-038 was a Phase 2, 26-week, randomized, double-blind, placebo-controlled, outpatient study in subjects with schizophrenia who had predominant negative symptoms while on adequate treatment with an antipsychotic. A total of 403 subjects were randomized to receive double-blind placebo (202 subjects) or pimavanserin (201 subjects) at 83 sites in North America and Europe, and 346 (85.9%) subjects completed the study (pimavanserin, 172 subjects [85.6%]; placebo, 174 subjects [86.1%]). Treatment began at 20 mg QD pimavanserin or matching placebo, could be adjusted to 10-34 mg QD between Weeks 2 and 8, and then remained stable.

Adding pimavanserin to existing antipsychotic treatment resulted in statistically significant improvement of negative symptoms of schizophrenia. A statistically significant improvement was observed in the pimavanserin group compared to the placebo group for the primary efficacy endpoint, the change from Baseline to Week 26 in the NSA-16 total score (p=0.0434). Improvement was observed in the pimavanserin group versus placebo at each postbaseline visit, achieving statistical significance at Week 4 (p=0.0334) and Week 20 (p=0.0067) as well as Week 26. In the post hoc analysis, significant superiority in the NSA-16 total score versus placebo was seen in pimavanserin subjects (56.9%) whose last dose level was 34 mg (p=0.0065), but not in subjects whose last dose level was 20 mg.

Statistically significant improvement, at the nominal alpha level of 0.05, in NSA-16 total score was observed in the pimavanserin group compared to the placebo group for subjects who were enrolled in Europe (p=0.0266), male (p=0.0016), White (p=0.0405), had a baseline body mass index (BMI) <25 kg/m<sup>2</sup> (p=0.0356), had schizophrenia duration >5 years (p=0.0009), had a duration of negative symptoms of schizophrenia >5 years (p=0.0005), or were markedly or severely ill, as defined by Clinical Global Impression Schizophrenia Scale-Severity (CGI-SCH-S) of negative symptoms score  $\geq 5$  (p=0.0199). Related clinical subgroups showed a similar magnitude of treatment effects for pimavanserin, but differences between treatment arms were smaller. However, the lack of separation was largely driven by higher responses in the placebo treatment group.

At Week 26, more subjects in the pimavanserin group compared to placebo were responders, based on percentage improvement on NSA-16 total score (46.7% vs. 41.8% of subjects with ≥20% improvement and 28.1% vs. 25.4% of subjects with ≥30% improvement). The change in NSA-16 domain scores from Baseline to Week 26 was numerically greater in the pimavanserin group for each domain score, with statistically significant improvement in the social involvement domain (p=0.0111).

Final Version: 2.0 Date: 29 February 2024 Clinical Study Protocol Amendment 3-Consolidated

Overall, safety results demonstrated that pimavanserin was generally safe and well-tolerated in subjects with schizophrenia.

#### 1.3.2 Phase 1 Study in Adolescents With Psychiatric Disorders

The PK profile of pimavanserin was evaluated in a Phase 1, open-label, multiple ascending dose (10, 20, or 34 mg) study in adolescents (male or female adolescents between 13 and <18 years) with psychiatric disorders (ACP-103-050). When adjusted for weight at Baseline, pimavanserin steady state systemic exposure was approximately dose proportional over the studied dose range (10 to 34 mg). There were no consistent differences in pimavanserin or N-desmethylpimavanserin, major metabolite of pimavanserin (AC-279) C<sub>max-ss</sub> and AUC<sub>τ</sub> between the age subsets; however, small differences observed were likely due to weight and not age. Accumulation of pimavanserin (approximately 3- to 5-fold overall) and AC-279 (approximately 13- to 18-fold) is consistent with adults and was expected based on the known respective half-lives (57 hours and 200 hours) relative to dosing interval. The parent (pimavanserin) to metabolite (AC-279) steady state ratio for  $C_{max-ss}$  and  $AUC_{\tau}$  was comparable across dose cohorts and ranged from 120% to 151%. These values are comparable to those in adults confirming the lack of difference in metabolism between adults and adolescents.

Additional information on previous pimavanserin clinical studies is provided in the pimavanserin Investigator's Brochure and in the US package insert for NUPLAZID® (pimavanserin) for oral use.

#### 1.4 **Study Rationale**

Irritability associated with ASD is often caused by multiple underlying comorbid conditions, many of which are linked to serotonergic system dysfunction. Based on the efficacy of two approved antipsychotics with 5-HT<sub>2A</sub> antagonism (and inverse 5-HT<sub>2A</sub> agonism in case of risperidone) it is hypothesized that pimavanserin, a more selective 5-HT<sub>2A</sub> inverse agonist/antagonist, may be effective in the treatment of irritability and other ASD symptoms.

#### **Rationale for Study Design** 1.4.1

This protocol describes an open-label extension study to determine the long-term safety and tolerability of pimavanserin for the treatment of irritability associated with ASD. The study follows a 6-week, Phase 2, dose ranging, randomized, double-blind, placebo-controlled study in pediatric patients (5 through 17 years of age) with a diagnosis of ASD will evaluate the efficacy, safety, and tolerability of pimavanserin by dose level (high pimavanserin dose and low pimavanserin dose).

While the focus of the double-blind study is to assess the efficacy of selected doses of pimavanserin versus placebo, evaluate the overall clinical benefit in various symptom domains and functioning, and obtain short-term safety and tolerability data, the purpose of this open-label extension is to obtain long-term information on the safety and tolerability of pimavanserin in children and adolescents. Exploratory information about the sustained efficacy of pimavanserin will also be collected in the efficacy assessments throughout the study. The primary endpoint is treatment-emergent adverse events (TEAEs).

Examining pimavanserin long-term safety, tolerability, and efficacy is of critical importance to eventually help clinicians make an informed decision on pharmacotherapy for patients.

#### 1.4.2 Rationale for Dose Selection

Selection of the pimavanserin high dose (34 mg for children and adolescents 13 through 17 years, and 20 mg for children 5 through 12 years) is based on achieving the same systemic exposure (maximum (peak) observed drug concentration [C<sub>max</sub>] and area under the plasma concentration-time curve [AUC]) in adults with pimavanserin 34 mg once daily that consistently demonstrated efficacy and safety in the adult population in several psychiatric conditions. Specifically, data from studies in Parkinson's disease psychosis, dementia-related psychosis, major depressive disorder, and schizophrenia, show that pimavanserin 34 mg QD is the more effective dose for adults. Similarly, exposure-response analyses consistently demonstrated that higher pimavanserin exposure is associated with greater response across all studied indications. Exposure associated with the 34 mg dose in adults was thus considered the "target exposure".

Stochastic simulations using actual and virtual adolescent (13 through 17 years) and adult populations (18 through 49 years) were undertaken to help guide pimavanserin dose selection in pediatric subjects within the age range of 5 through 17 years (ACP-103-MS-010) that are likely to achieve the target exposure. The results showed that compared to the adult population (18 through 49 years), steady-state AUC for the 34 mg dose was largely consistent across all age groups (5 through 49 years) and body weight groups (16 through >75 kg) with comparable median values and considerable overlap in the distribution of AUC values across the different groups.

Steady state C<sub>max</sub>, following 34 mg dosing, was progressively higher with decreasing age, as well as with decreasing body weight. A 20 mg dose produced C<sub>max</sub> exposures in children 5 through 9 years of age that were comparable to the 34 mg dose in the adolescents and adults. Because body-weight adjusted PK for children 12 years and younger are usually different from adolescents and adults for similar doses, a conservative approach was adopted and the older children (10 through 12 years) were grouped with the younger children (5 through 9) to receive the lower doses. As such, the selected high dose that achieves the target exposure (equivalent to a 34 mg dose in adults) for children 5 through 12 years is 20 mg. For children and adolescents 13 through 17 years the selected dose is 34 mg to achieve the target exposure


The pimavanserin low dose (20 mg for children and adolescents 13 through 17 years of age, and 10 mg for children 5 through 12 years of age) was selected to reduce the extent of exposure overlap between the low and high dose, while offering the potential to explore efficacy in ASD patients with lower pimavanserin doses/exposures that were well tolerated in the adult population in various psychiatric indications.

### Rationale for dosing periods

To ensure safe rollover of those subjects previously on placebo and minimize the risks of potential unblinding all eligible subjects will receive pimavanserin "low dose" for the first two weeks of the study. Subjects who were on "old dose" during the antecedent double-blind study will likely experience ccl efficacy during this period, due to the long half-life of pimavanserin, and having achieved steady state by the end of the antecedent double-blind study. At the Week 2 visit, the dose may be increased to pimavanserin "high dose", based on the Investigator's assessment of clinical response.

After the Week 2 visit, and up to and including the Week 20 visit, dose adjustments, either increases or decreases, may be made at any clinic visit (scheduled or unscheduled), based on the Investigator's assessment of clinical response and tolerability.

No further dose adjustments are allowed after the Week 20 visit.

#### 1.5 **Benefit/Risk Assessment**

#### 1.5.1 **Known Potential Risks**

The Prescribing Information for NUPLAZID® (pimavanserin) tablets and capsules for oral use (Acadia Pharmaceuticals Inc. 2020) includes the following Boxed Warning:

"WARNING: INCREASED MORTALITY IN ELDERLY PATIENTS WITH **DEMENTIA-RELATED PSYCHOSIS"** 

The increased mortality warning in elderly patients with dementia-related psychosis is based on information regarding antipsychotic drugs in general, rather than specific pimavanserin data.

The Warnings and Precautions section of the Prescribing Information for pimavanserin also includes information about QT interval on ECG (QT) interval prolongation. Pimavanserin prolongs the QT interval. The use of pimavanserin should be avoided in patients with known QT prolongation or in combination with other drugs known to prolong QT interval including Class 1A antiarrhythmics (e.g., quinidine, procainamide) or Class 3 antiarrhythmics (e.g., amiodarone, sotalol), certain antipsychotic medications (e.g., ziprasidone, chlorpromazine, thioridazine), and certain antibiotics (e.g., gatifloxacin, moxifloxacin). Pimavanserin should also be avoided in patients with a history of cardiac arrhythmias, as well as other circumstances that may increase the risk of the occurrence of torsade de pointes and/or sudden death, including

prolongation of the QT interval.

symptomatic bradycardia, hypokalemia or hypomagnesemia, and the presence of congenital

NUPLAZID is contraindicated in patients with a history of a hypersensitivity reaction to pimavanserin or any of its components. Rash, urticaria, reactions consistent with angioedema (e.g., tongue swelling, circumoral edema, throat tightness, and dyspnea) have been reported. In addition, adverse reactions of somnolence, falls, agitation, and aggression have been reported during postapproval use of NUPLAZID.

Pimavanserin has not yet been studied as monotherapy in children and adolescents therefore no data are available on specific risks in this population. In adolescents treated with pimavanserin in combination with other psychotropics, pimavanserin dose-related QTc prolongation, and a trend for higher exposure with decreasing age and decreasing body weight, have been observed.

### 1.5.2 Known Potential Benefits

Pimavanserin has not been studied in children and adolescents with ASD, thus there are no known benefits. It has shown antipsychotic properties in the indications of PDP, and is currently being evaluated as adjunctive treatment in adults with negative symptoms of schizophrenia. Based on the mechanism of action of pimavanserin, potential benefits may include its clinical utility in the treatment of irritability and other symptoms of ASD. This is particularly the case with subjects previously randomized to placebo. Subjects may benefit from the increased medical care and attention for the study duration.

A detailed summary of the potential risks and benefits is available in the pimavanserin Investigator's Brochure.

### 2 STUDY OBJECTIVES AND ENDPOINTS

### 2.1 Primary Objective

• To evaluate the long-term safety and tolerability of pimavanserin after 52 weeks of treatment in children and adolescents with ASD

### 2.1.1 Primary Endpoints

• Treatment-emergent adverse events (TEAEs)

Safety will also be evaluated by analyses of the following:

- Vital signs
- Weight and body mass index (BMI)
- 12-lead electrocardiograms (ECGs)
- Physical examination results


- Clinical laboratory tests (including urinalysis) and hormonal assessments
- Columbia—Suicide Severity Rating Scale (C-SSRS)
- Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A)

#### 2.2 **Secondary Objective**

• To evaluate the continued response to long-term pimavanserin treatment in children and adolescents with ASD

#### 2.2.1 **Secondary Endpoint**

• Proportion of subjects who have at least 25% reduction from the antecedent study Baseline in the Aberrant Behavior Checklist-Irritability (ABC-I) subscale score AND a Clinical Global Impression–Improvement (CGI-I) of irritability score of 1 (very much improved) or 2 (much improved) compared to the antecedent study baseline status at Week 52.

#### 2.3 **Exploratory Objectives**

- To evaluate the continued benefit of long-term pimavanserin treatment on the symptoms of ASD, in children and adolescents with ASD in the following clinical areas:
  - o Aberrant Behavior Checklist (ABC) symptom domains
  - Maintenance of benefit
  - Response to treatment

#### 2.3.1 **Exploratory Endpoints**

- Change from Baseline at Week 52 in the caregiver-rated ABC subscale scores:
  - Irritability
  - Stereotypic behavior
  - Lethargy
  - Hyperactivity
  - Inappropriate speech
- Change from Baseline at Week 52 in the Clinical Global Impression—Severity (CGI-S) of irritability score
- CGI-I of irritability score from the antecedent study Baseline at Week 52
- Change from Baseline at Week 52 in the Caregiver Strain Questionnaire (CGSQ)
- Proportion of subjects who have at least 25% reduction from the antecedent study Baseline in the ABC-I subscale score (ABC-I responders) at Week 52


• Proportion of subjects who have CGI-I of irritability score of 1 (very much improved) or 2 (much improved) compared to the antecedent study baseline status (CGI-I of irritability responders) at Week 52

### STUDY DESCRIPTION

#### 3.1 **Overview of Study Design**

This study will be conducted as a 52-week, open-label extension study of the antecedent double-blind study to determine the long-term safety and tolerability of pimavanserin for the treatment of irritability associated with ASD in children and adolescents (5 through 17 years old at the time of enrolling into the antecedent double-blind study). Approximately 60 global sites and approximately eight countries will participate in this study.

The duration of participation for individual study subjects will be up to approximately 56 weeks. The total duration of exposure to pimavanserin may be greater than 52 weeks (e.g., up to 58 weeks) as some subjects have been treated with pimavanserin in an antecedent double-blind study.

The study will have two periods:

- Open-label treatment period (52 weeks)
- Safety follow-up period (at least 30 days)

Subjects who have completed the antecedent double-blind study and who have shown no significant worsening of symptoms at the end of the study as evidenced by the CGI-I of irritability will be included in this long-term extension study.

Study ACP-103-070 subjects must be consented prior to the procedures being performed at the End of Treatment (EOT) visit in the antecedent double-blind study. Procedures performed at the EOT visit of the antecedent double-blind study will be carried over to the ACP-103-070 study to be included as baseline information, and this visit will be considered the Baseline Visit (Visit 1) of the ACP-103-070 study.

The study start date is defined as the date the first subject is enrolled, which is the baseline visit date for the first subject for this open-label study.

The primary completion date is the last date that subject data was collected for the primary outcome measure.

The study completion date (End of Study) is defined as the last date that subject data was collected, which includes the safety follow-up telephone call visit. Procedures for when a subject is lost to follow-up are provided in Section 4.6.

3.1.1 Open-label Treatment Period (52 Weeks)

## Subjects will be stratified by age group (5- through 12-year-olds or 13- through 17-year-olds). Subjects will remain in the age group they were stratified into during the antecedent double-blind

study, throughout the OLE study.

All subjects will receive QD doses of pimavanserin over 52 weeks of treatment. Subjects will start at the "low dose" for their age group (10 mg for 5- through 12-year-olds; 20 mg for 13- through 17-year-olds) for the first two weeks. At the Week 2 visit, the daily dose may be adjusted to the "high dose" for their age group (20 mg for 5- through 12-year-olds; 34 mg for 13- through 17-year-olds), based on the Investigator's assessment of clinical response. After the Week 2 visit and up to and including the Week 20 visit, dose adjustments, either increases or decreases, may be made at any clinic visit (scheduled or unscheduled), based on the Investigator's assessment of clinical response and tolerability. No further dose adjustments are allowed after the Week 20 visit.

During the treatment period, clinic visits will be conducted at Baseline and Weeks 2, 6, 12, 20, 28, 36, 44, and 52, or upon early termination (ET) from the study.

Study drug will be dispensed to the subject to take home at the Baseline visit and at each subsequent clinic visit. The subject and their parent/legally acceptable representative (LAR) will be provided instructions for the subject's first dose of study drug the day after the Baseline visit. It is recommended that the subject take the study drug at approximately the same time each day as a single, oral dose.

All concomitant medications should remain at a stable dose throughout the study, if possible, except as described in Appendix A to minimize confounding interpretation of any correlating pimavanserin dose changes, including treatment discontinuations.

### 3.1.2 Safety Follow-up Period (30 Days)

A follow-up safety assessment will be conducted by telephone call at least 30 days after the last dose of study drug. The safety follow-up assessment will not be done if the subject (and/or parent/LAR) withdraws consent to participate in all parts of the study.

### 4 SUBJECT ELIGIBILITY AND WITHDRAWAL CRITERIA

To be eligible for this study, subjects must meet all of the inclusion criteria and none of the exclusion criteria to enter this open-label extension study.


Study: ACP-103-070
Clinical Study Protocol Amendment 3-Consolidated

### 4.1 Inclusion Criteria

A subject must meet all of the following inclusion criteria to be eligible for participation in the study:

### Study Population

- 1. Has completed the treatment period of the antecedent double-blind study
- 2. Informed consent prior to the conduct of any study procedures is required as follows:
  - a. The subject should provide written or oral assent if deemed able by the Investigator.
  - b. The subject's parent/LAR must provide written consent. The subject's parent/LAR must be considered reliable by the Investigator, able to complete assessments regarding the subject's development and behavior throughout the study, and able to help ensure compliance with study treatment, study visits, and protocol procedures.
  - c. If a person other than the parent/LAR has been designated as a caregiver for the purpose of providing input for caregiver-reported scales, that person must also provide written consent. Such a designee should be a family member, adult and responsible, living with or in very frequent contact with the subject participating in the study, who is committed to providing responses for the caregiver-reported scales for the duration of the study.

The process of obtaining informed consent will be conducted in accordance with institutional review board (IRB) or ethics committee (EC) policy and applicable local law

3. In the Investigator's opinion, the subject, to the best of his/her ability, the parent/LAR, and the designated caregiver (if applicable, and in accordance with IRB or EC policy and applicable local law) are able to understand the nature of the study, follow protocol requirements and be willing to comply with study drug administration requirements

### Psychiatric Diagnosis

- 4. Continues to be both clinically stable and not at imminent risk of suicide or injury to self, others, or property, in the opinion of the Investigator
- 5. Continues to be medically stable at enrollment, in the opinion of the Investigator


Study: ACP-103-070 Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

### **Contraceptives**

6. Female subjects who participate in this study must either be unable to become pregnant (e.g., premenarchal, surgically sterile, etc.) -OR- must agree to use two clinically acceptable methods of contraception (e.g., oral, intrauterine device [IUD], diaphragm plus spermicide, injectable, transdermal or implantable contraception) during the treatment period, and for at least 45 days after last dose.

All female subjects of childbearing potential must have a negative urine human chorionic gonadotropin (hCG) pregnancy test at Baseline and all clinic visits. Females of childbearing potential are defined as females who have begun menstruating.

### 4.2 Exclusion Criteria

A subject must meet none of the following exclusion criteria to be eligible for the study:

### Study Population

1. Subject or parent/LAR is judged by the Investigator to be inappropriate for the study (e.g., significantly noncompliant in the antecedent double-blind study)

### CNS, Psychiatric, and Illicit Drug Use Criteria

- 2. Requires treatment with a medication prohibited by the protocol, including concomitant psychotropic drugs targeting irritability, including those used off-label (clonidine, guanfacine, and propranolol; lithium, valproate), medications that prolong the QT interval; and strong cytochrome P450 (CYP) 3A4 enzyme (CYP3A4) inhibitors and inducers (see Appendix A and Appendix B)
- 3. Is at a significant risk of suicide, or is a danger to self or others, in the opinion of the Investigator based upon all available sources of information including C-SSRS (positive answer to suicidal ideation questions 4 or 5 [or positive answer to suicidal behavior questions at Baseline])
- 4. Is at risk of significant violent behavior to the extent that participation would pose an undue risk to other patients, caregivers, or others in the opinion of the Investigator
- 5. Has a positive urine drug test at Baseline. For study eligibility, the urine toxicology (drug) screen (UDS) must be negative for any substance for which the subject does not have a valid prescription.

Study: ACP-103-070 Clinical Study Protocol Amendment 3-Consolidated

Medical Criteria

# 6. Has developed a serious and/or unstable psychiatric, neurologic, cardiovascular (e.g., long QT syndrome, torsade de pointes, unstable cardiac syndrome or syncope, congestive heart failure, ongoing uncorrected hypokalemia or hypomagnesemia, non-sustained or sustained

- ventricular tachycardia), respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies that, in the judgment of the Investigator, would jeopardize the safe participation of the subject in the study, or has major surgery planned during the study
- 7. Has experienced any change in medical or treatment status that may increase the risk
- associated with taking pimavanserin, would interfere with safety assessments, or would confound the interpretation of study results, based on the Investigator's judgment
- 8. For age <13 years, a resting position (sitting or supine) systolic (SBP) and/or diastolic blood pressure (DBP) level ≥90th percentile for gender-specific age and height charts from the National Heart and Lung Institute (NHLI), at Baseline. For age ≥13 years a resting position (sitting or supine) SBP ≥120 mmHg and/or a DBP ≥80 mmHg, at Baseline.
- 9. Has a clinically significant abnormal ECG at Baseline or any of the following cardiac conduction abnormalities:
  - a. Corrected QT interval using Fridericia's correction method (QTcF) ≥450 ms
  - b. PR interval on ECG >220 ms
  - c. Evidence of second- or third-degree atrioventricular block
  - d. Evidence of complete left bundle branch block
  - e. Intraventricular conduction delay with QRS interval on ECG (QRS) >110 ms
  - f. QRS or T wave morphology that could, in the Investigator's opinion, render QT interval assessment unreliable
  - g. Sick sinus syndrome
  - h. Non-sinus rhythm
  - i. Resting heart rate <50 beats per minute

One repeat set of triplicate ECGs is allowed at Baseline.

- 10. Weight <15 kg
- 11. *In Italy only*: Has a sensitivity to any compound present in pimavanserin or any metabolites or compounds listed in the Investigator's brochure as being present in this medication


#### 4.3 Screen Failures

The Investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

#### 4.4 **Subject Withdrawal of Consent**

In accordance with the Declaration of Helsinki and other applicable regulations, a subject has the right to withdraw from the study at any time, and for any reason, without prejudice to his or her future medical care.

If the subject (and/or parent/LAR) decides to withdraw consent from all components in the study, this must be documented and no additional assessments will be performed. The Sponsor may retain and continue to use any data collected before such a withdrawal of consent. The subject may request destruction of any samples taken and not tested, prior to their withdrawal of consent, and the Investigator must document this in the site study records.

If the subject (and/or parent/LAR) wants to discontinue treatment and agrees to the evaluations specified at the EOT/ET visit and/or at safety follow up (whichever is applicable), as outlined in Table S-1, the agreed assessments should be conducted. The subject's reason for wanting to discontinue treatment and the agreement to continue with the applicable assessments for study termination must be documented.

Every reasonable effort should be made to keep the same parent/LAR or designee who completed the observer's study scales in study ACP-103-069 to complete them throughout study ACP-103-070 in order to maintain the validity of the scoring.

#### 4.5 **Subject Discontinuation**

Subjects may be discontinued from the study treatment for a number of reasons, including, but not limited to, those listed below:

- Adverse event
- Death
- Lack of efficacy
- Lost to follow-up (Section 4.6)
- Non-compliance with study drug
- Physician decision
- Pregnancy
- Protocol deviation

Study: ACP-103-070 Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

- Study terminated by sponsor
- Use of prohibited medication
- Withdrawal of consent by subject (or by parent/LAR)
- Other

### 4.5.1 Handling of Subject Discontinuation During the Treatment Period

Unless the subject (or parent/LAR) has withdrawn consent from all components of the study, every reasonable effort should be made to complete Visit 6/ET and the safety follow-up visit (as outlined in Table S-1) if a subject discontinues prematurely during the treatment period of the study. All information will be reported on the applicable pages of the electronic case report form (eCRF).

If a subject is discontinued from the study treatment because of an AE, every reasonable attempt should be made to follow and appropriately treat (or refer for treatment) the subject until the AE resolves or until the Investigator deems the AE to be chronic or stable. For subjects who continue to be followed for safety, serious adverse events (SAEs) should continue to be reported as described in Section 7.4.2. All SAEs will continue to be followed and appropriately treated until such events have resolved or the Investigator deems them to be chronic or stable.

### 4.6 Subject Lost to Follow-up

A subject will be considered lost to follow-up if they fail to attend a scheduled visit (including the safety follow-up visit) and the study subject or parent/LAR is unable to be contacted by the study site **after repeated attempts**.

Every reasonable effort should be made to contact the subject and parent/LAR and will include a minimum of three documented phone calls and, if necessary, a certified letter to the subject's last known mailing address or local equivalent methods. All contact attempts are to be documented in the source documents.

### 4.7 Study Discontinuation

The Sponsor reserves the right to discontinue the study at any time for any reason. Such reasons may be any of, but not limited to, the following:

- Occurrence of AEs unknown to date in respect of their nature, severity, and duration or the unexpected incidence of known AEs
- Medical, ethical, or business reasons affecting the continued performance of the study

Regulatory authorities also have the right to terminate the conduct of the study in their region for any reason.

### 4.8 Prior and Concomitant Therapy

All medications used from study baseline until completion of the safety follow-up visit are to be recorded.

### 4.8.1 Prior Medication

Prior medication is defined as any medication with a stop date prior to the date of the first dose of study drug.

### 4.8.2 Concomitant Medication

Concomitant medication is defined as any medication that is ongoing at the first dose of study drug or with a start date between the dates of the first dose and last dose of study drug, inclusive.

In order to ensure that appropriate concomitant therapy is administered, it is essential that subjects be instructed not to take any medication without prior consultation with the Investigator (unless the subject is receiving treatment for a medical emergency). Non-pharmacological treatment should remain the same throughout the study duration.

The Investigator may prescribe appropriate medication to treat AEs (see Appendix A and Appendix B).

### 4.8.2.1 Permitted, Restricted, and Prohibited Medications

Prohibitions and restrictions for concomitant medications should be followed between the Baseline visit and Visit 6/EOT/ET as specified in Appendix A and Appendix B. These appendices do not constitute an exhaustive list and any questions regarding prohibited and restricted medications should be discussed with the Medical Monitor or designee. The Investigator may prescribe appropriate medication to treat AEs.

Medications that can prolong QT interval are prohibited (or restricted) as specified in Appendix A.

Permitted concomitant medications should remain at a stable dose throughout the treatment period.

If a subject is on a medication restricted by the protocol, the medication should be adjusted if it is determined by the Investigator to be clinically appropriate (e.g., if the subject's symptoms are not well-controlled or if the subject cannot tolerate the current medication) in consultation with the treating physician.

Subjects who require current treatment with a prohibited medication will be withdrawn from the study.

Subjects who have taken a prohibited medication during the study will be withdrawn from the study unless:

- the prohibited medication has been discontinued, AND
- withdrawal from the study presents an unacceptable medical risk to the subject

The justification to allow the subject who has taken a prohibited medication to continue in the trial will be made by the Sponsor/Medical Monitor, with medical input from the Investigator, and will be documented. If a subject is allowed to remain in the trial, this will be reported as a major protocol deviation and not a waiver.

### 4.8.3 Rescue Medications, Treatments, and Procedures

Rescue medication, as determined by the Investigator, is permitted for a maximum of 7 consecutive days, provided it is consistent with the prohibitions and restrictions in Appendix A and Appendix B.

### 5 INVESTIGATIONAL PRODUCT

### 5.1 Investigational Product Description

The investigational product will be pimavanserin 10 mg (provided as  $1\times10$  mg capsule), pimavanserin 20 mg (provided as  $1\times20$  mg capsule), or pimavanserin 34 mg (provided as  $1\times34$  mg capsule). Capsules will be administered orally as a single dose once daily.

Pimavanserin dosages below:

Pimavanserin 10 mg (provided as 1×10 mg capsule)

Pimavanserin 20 mg (provided as 1×20 mg capsule)

Pimavanserin 34 mg (provided as 1×34 mg capsule)

### 5.1.1 Formulation, Appearance, Packaging, and Labeling

The Sponsor will supply pimavanserin 10 mg, 20 mg and 34 mg capsules.

Pimavanserin 10 mg, 20 mg, and 34 mg capsules, are white to off-white capsules.

Each 34 mg pimavanserin capsule contains 40 mg of pimavanserin tartrate, which is equivalent to 34 mg of pimavanserin free base.

Each 20 mg pimavanserin capsule contains 23.5 mg of pimavanserin tartrate, which is equivalent to 20 mg of pimavanserin free base.

Each 10 mg pimavanserin capsule contains 11.8 mg of pimavanserin tartrate, which is equivalent to 10 mg of pimavanserin free base.


Inactive ingredients include magnesium stearate, microcrystalline cellulose, and the components of the capsule shell (hypromellose and titanium dioxide).

Pimavanserin capsules are manufactured under current Good Manufacturing Practice.

Pimavanserin capsules will be provided in kits containing two blister cards, with each card containing 10 capsules in a blister strip (total 20 capsules per kit). Each kit will be labeled as required per country requirement.

During the treatment period, study drug will be distributed in a quantity sufficient to ensure the subject has an adequate supply of study drug between study visits.

#### 5.1.2 **Product Storage and Stability**

Investigational product must be stored in a secure area with restricted access, not above 25°C (77°F), and according to local and national regulations. To prevent potential capsule color fading, protect from light.

#### 5.1.3 **Dosing and Administration**

At the Baseline visit of Study ACP-103-070, study drug will be dispensed to the subject to take home. The subject and their parent/LAR will be provided instructions for the subject's first dose of study drug on the day after the Baseline visit.

Each daily dose consists of one capsule. Subjects should be instructed to take one capsule, orally, once daily, in the morning, at the same time every day. Subjects should be instructed to not to open the capsules. The capsules may be taken with or without food.

#### 5.1.3.1 **Dose Modification**

All subjects will receive the "low dose" for their age group for the first two weeks of the study. After the Week 2 visit the dose may be increased to the "high dose" based on the Investigator's assessment of clinical response. After the Week 2 visit, and up to and including the Week 20 visit, dose adjustments, either increases or decreases, may be made at any clinic visit (scheduled or unscheduled), based on the Investigator's assessment of clinical response and tolerability.

No further dose adjustments are allowed after the Week 20 visit.

#### 5.1.4 Blinding

This is an open-label study.

#### 5.1.5 **Study Drug Compliance**

The Investigator or designated study center personnel will maintain a log of all study drug dispensed and returned during the study. Study drug supplies for each subject will be inventoried and accounted for throughout the study to verify the subject's compliance with the dosage regimen. Subjects will be counseled regarding compliance at every visit. Subjects who have <80% or >120% compliance may be discontinued from the study. If a subject shows significant undercompliance (<80%) between any two scheduled visits, the Medical Monitor should be notified to determine if the subject remains eligible for the study and whether the incident should be considered a protocol deviation.

If a subject misses one dose of study drug, he or she should not take an extra dose the next day.

### 5.1.6 Overdose

An overdose is a deliberate or inadvertent administration of a treatment at a dose higher than the maximum recommended dose per protocol. It must be reported using the Sponsor's Overdose Reporting form, irrespective of outcome, even if toxic effects were not observed (Section 7.4.4). All events of overdose are to be captured as protocol deviations.

### 5.2 Investigational Product Accountability Procedures

The Investigator or designee will keep current and accurate records of the study drug product dispensed, used, and returned for each subject to assure the regulatory authority and the Sponsor that the study drug is being handled appropriately. Subjects should be instructed to return all packaging and unused study drug to the Investigator at regularly scheduled clinic visits and ET visits. Any study drug supplied is for use in this study only and should not be used for any other purpose.

At appropriate intervals during the study, study drug reconciliation will be performed by the Sponsor (or designee) who may return appropriate unused study drug and used and unused packaging to the Sponsor's designee for destruction.

At the conclusion of the study, final study drug reconciliation will be conducted at the site. Final study drug accountability documentation will be maintained at both the site and at the Sponsor. Any remaining unused study drug and all used and unused packaging will be sent back to the Sponsor's designee for destruction, as allowed by country specific regulations. Documentation of study drug destruction will be recorded and maintained by both the Sponsor and the Sponsor's designee.

### **6 STUDY ASSESSMENTS**

Study specific assessments are detailed below. All assessments will be completed according to the schedule described in Table S-1. Every effort should be made to complete the required procedures and evaluations at the designated visits and times.

For scales that require caregiver input, the caregiver should be the parent/LAR or designee. A designee should be a family member, adult and responsible, living with or in very frequent


contact with the subject participating in the study, who is committed to providing responses for the caregiver-reported scales for the duration of Studies ACP-103-069 and ACP-103-070. Caregivers providing input for the ABC, RBS-R, and CGSQ scales will be trained in accurate symptom reporting (ASR) prior to completing the scales. ASR training should be done at Screening in the antecedent study (Study ACP-103-069) before the caregiver completes any

scales, and repeated whenever there is a change in caregiver or if the site feels a caregiver

### **6.1** Baseline Assessments

requires retraining.

Subject consent for the present study must be obtained prior to the final procedures being performed at the EOT visit of the antecedent double-blind study and before any new procedures are performed for Study ACP-103-070. Data from the EOT procedures of antecedent double-blind study will be carried over to the ACP-103-070 study to be included as baseline information for the present study and this visit will be considered Baseline (Visit 1). Subject eligibility will be assessed by the site and the Sponsor through an eligibility review process.

### 6.1.1 Physical Examination and Self- or Caregiver-reported Tanner Staging

See Section 6.4.1

### 6.1.2 Vital Signs

See Section 6.4.2.

### 6.1.3 Height, Weight, and Body Mass Index

See Section 6.4.1.

### 6.1.4 12-lead ECG

See Section 6.4.3.

### **6.1.5** Clinical Laboratory Tests

See Section 6.4.4.

### 6.1.6 Pregnancy Test

See Section 6.4.4.

### 6.1.7 Urine Toxicology (Drug) Screen

See Section 6.4.4

### **6.1.8** Aberrant Behavior Checklist

See Section 6.2.1.


Study: ACP-103-070 Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

### 6.1.9 **CGI-S**

See Section 6.2.2.

### 6.1.10 CGI-I

See Section 6.2.3

### 6.1.11 RBS-R

See Section 6.2.4.

### 6.1.12 VABS-Socialization

See Section 6.2.5.

### 6.1.13 CGSQ

See Section 6.2.6.

### 6.1.14 C-SSRS

See Section 6.3.1

### 6.1.15 ESRS-A

See Section 6.3.2

### **6.1.16** Concomitant Medications and Adverse Events

All medications used from Baseline until completion of the safety follow up visit are to be recorded (Section 4.8).

All adverse events (Section 7) from Baseline until completion of the safety follow up visit are to be recorded.

### **6.2** Efficacy Assessments

### **6.2.1** Aberrant Behavior Checklist

The Aberrant Behavior Checklist (ABC) is a caregiver-rated scale comprised of five empirically-derived subscales encompassing 58 items that describe various behavior problems (Aman et al. 1985; Kaat et al. 2014). The subscales have been labeled:

- I. Irritability (irritability, agitation, and crying) (15 items)
- II. Lethargy (lethargy and social withdrawal) (16 items)
- III. Stereotypic Behavior (7 items)
- IV. Hyperactivity (hyperactivity and noncompliance) (16 items)
- V. Inappropriate Speech (4 items)

The ABC will be administered at Baseline, and at all visits from Week 2 through Week 52. A score for each item ranges from 0 indicating "not at all a problem" to 3 indicating "the problem is severe in degree". Subscale scores are calculated by summing the items within that subscale. Higher scores indicate greater impairment.

The reliable caregiver identified upon subject's ACP-103-070 Baseline visit will complete the rating scale. A clinician will be available to assist the caregiver during completion of the questionnaire.

This assessment will take approximately 10 to 20 minutes to complete.

The same rater or clinician should perform the ABC throughout the study together with the same caregiver as established at the Baseline visit.

### 6.2.2 CGI-S

The CGI-S is a clinician-rated, 7-point scale that is designed to rate the severity of the subject's illness, in this case irritability associated with ASD, at the time of assessment, making use of the clinician's judgment and past experience with subjects who have the same disorder (Guy 1976). The CGI-S of irritability will be administered at Baseline, and at all visits from Week 2 through Week 52. The same clinician should administer the CGI-S of irritability throughout the study as established at the Baseline visit.

### 6.2.3 CGI-I

The CGI-I is a clinician-rated, 7-point scale that is designed to assess how much the subject's illness, in this case irritability associated with ASD, has improved or worsened relative to a baseline state at the beginning of the intervention (Guy 1976). In this study, improvement or worsening is assessed relative to the baseline status in the antecedent double-blind study.

The CGI-I of irritability will be administered at Baseline, and at all visits from Week 2 through Week 52.

The same clinician should administer the CGI-I of irritability throughout the study as established at the Baseline visit.

### 6.2.4 Repetitive Behavior Scale–Revised

The Repetitive Behavior Scale–Revised (RBS-R) (Lam and Aman 2007) is a 43-item parent/caregiver-facing questionnaire. Items are conceptually grouped into six subscales:

- stereotyped behavior (movements with no obvious purpose that are repeated in a similar manner)
- self-injurious behavior (actions that cause or have the potential to cause redness, bruising, or other injury to the body)


Final Version: 2.0 Date: 29 February 2024 Clinical Study Protocol Amendment 3-Consolidated

- compulsive behavior (behavior that is repeated and performed according to a rule or involves things being done "just so")
- ritualistic behavior (performing activities of daily living in a similar manner)
- sameness behavior (resistance to change, insisting that things stay the same)
- restricted behavior (limited range of focus, interest, or activity)

Items are rated on a 4-point Likert scale ranging from (0) "behavior does not occur" to (3) "behavior occurs and is a severe problem", and raters are asked to refer to the previous month when completing the scale.

The RBS-R will be administered at Baseline, and at the Week 12, Week 28, Week 36, Week 44, and Week 52 visits. This scale will take approximately 20 to 30 minutes to complete.

The same rater or clinician should perform the RBS-R throughout the study together with the same caregiver as established at the Baseline visit.

#### 6.2.5 **Vineland Adaptive Behavior Scales-Socialization**

The Vineland Adaptive Behavior Scales (VABS) is a parent/caregiver-facing measure of adaptive behavior, organized into three domains: communication, daily living skills, and socialization (Sparrow et al. 2016). Only the socialization domain will be used in this study.

The VABS-Socialization will be administered at Baseline, and at the Week 12, Week 28, Week 36, Week 44, and Week 52 visits.

The same rater or clinician should perform the VABS-Socialization together with the same caregiver throughout the study as established at baseline visit.

#### 6.2.6 **Caregiver Strain Questionnaire**

The CGSQ (Brannan et al. 1997) is a 21-item parent/caregiver-facing questionnaire of self-reported strain experienced since last visit by parents/caregivers and families of youth with emotional problems. Responses are on a 5-point Likert scale ranging from (1) "not at all a problem" to (5) "very much a problem".

The following areas of strain are included:

- disruption of family life and relationships
- demands on time
- negative mental and physical health effects for any member
- financial strain
- sacrifice

Study: ACP-103-070 Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

- disruption of social/community life
- worry and guilt
- fatigue and strain
- embarrassment
- child-caregiver relationship

The CGSQ will be administered at Baseline, and at the Week 6, Week 20, Week 28, Week 36, Week 44, and Week 52 visits.

The same rater or clinician should perform the CGSQ together with the same caregiver throughout the study as established at Baseline visit.

### 6.3 Safety Scales

### 6.3.1 Columbia-Suicide Severity Rating Scale

The C-SSRS monitors changes in suicidal thinking and behavior over time, in order to determine risk (Posner et al. 2011). The following four constructs are measured: the severity of ideation, the intensity of ideation, behavior, and lethality.

The C-SSRS will be used to assess suicidal ideations and behaviors; the Since Last Visit version will be administered at Baseline, and at all subsequent visits. The C-SSRS results for each subject should be reviewed by the Investigator at each visit. If at any time the C-SSRS results for a given subject reveal potential suicidality, then the Investigator should assess the clinical significance of such results. If a clinically significant risk of suicidality is identified for a subject, then the Investigator should discontinue the subject and implement appropriate treatment (Sections 4.4 and 3.1.2).

The C-SSRS will be administered at Baseline, at all visits from Week 2 through Week 52, and at unscheduled visits.

The same rater or clinician should perform the C-SSRS together with the same caregiver throughout the study as established at Baseline visit.

### 6.3.2 Extrapyramidal Symptom Rating Scale-Abbreviated

The ESRS (Chouinard and Margolese 2005) was developed to assess drug induced movement disorders such as parkinsonism, akathisia, dystonia and tardive dyskinesia with established reliability, validity, and sensitivity. It consists of a questionnaire of parkinsonian symptoms, physician examination of parkinsonism, dyskinetic movements, and global impression of tardive dyskinesia. The ESRS-A, an accepted modified form of the original ESRS, will be used during


the study to monitor for any worsening in extrapyramidal symptoms or signs at scheduled and unscheduled visits.

The ESRS-A will be administered at Baseline, at all visits from Week 2 through Week 52, and at unscheduled visits.

The same rater or clinician should perform the ESRS-A together with the same caregiver throughout the study as established at Baseline visit.

#### 6.4 **Safety Assessments**

As known potential class side effects of antipsychotics, the following adverse events will be actively monitored, including hyperglycemia, leucopenia/neutropenia/agranulocytosis, orthostatic hypotension/bradycardia/syncope, QTc prolongation, akathisia and other extrapyramidal symptoms, weight gain, and somnolence. Criteria for identifying potentially clinically important laboratory values, ECG values, and vital signs are presented in Appendix C, Appendix D, and Appendix F, respectively; and criteria for identifying additional ECG measurements of potential clinical relevance for Medical Monitoring purposes are presented in Appendix E.

Circumstances may arise (e.g., pandemic, natural disaster, political upheaval, or technical issues) when on-site assessments of safety measures may not be possible. In those cases, assessments may be performed at the subject's place of residence either in person or via video technology or telephone, where possible. If a subject is unable to come to the site for lab draws and the site is unable to travel to the subject's place of residence, the subject may visit a local lab to obtain all safety labs. The Investigator must contact the Medical Monitor for approval with the plan. Sites must keep a log to identify details of all visits that are administered remotely.

#### 6.4.1 Physical Examination and Self- or Caregiver-reported Tanner Staging

A general physical examination will be conducted.

Height will be measured and reported.

Weight will be measured and reported.

Body mass index will be calculated using the following formula:

Weight  $(kg) / [height (m)]^2$ .

Tanner staging is a scale of physical development in children, adolescents, and adults. The scale defines physical measurements of development based on external primary and secondary sex characteristics, such as the size of the breasts, genitals, testicular volume and development of pubic hair (Marshall and Tanner 1969; Marshall and Tanner 1970).

Clinical Study Protocol Amendment 3-Consolidated

Date: 29 February 2024

A physical examination will be administered, and Tanner staging will be reported (either by the subject or the subject's caregiver), at Baseline, and at the Week 12, Week 28, Week 44, and

Week 52 visits.

Height (as measured by a stadiometer), weight, and BMI will be measured at Baseline, at all visits from Week 2 through Week 52, and at unscheduled visits.

### 6.4.2 Vital Signs

Vital signs will include body temperature, resting respiration rate, sitting (or supine) systolic and diastolic blood pressure, and pulse rate. The sitting (or supine) blood pressure should be measured after the subject has been sitting (or supine) for ≥3 minutes. If the initial blood pressure measurement is:

- ≥90th percentile systolic and/or diastolic for gender-specific age and height charts from the National Heart and Lung Institute (NHLI) for subjects under 13 years or
- ≥120 mmHg systolic or ≥80 mmHg diastolic for subjects 13 through 17 years,

at least 5 minutes rest should be allowed after the first measurement; then two additional blood pressure measurements are to be performed consecutively. The average of the three blood pressure measurements, systolic and diastolic, is the final blood pressure measurement and this average is the one to be entered into the EDC. All of the three blood pressure measurements with documentation of the time starting the resting and the time at which the two additional blood pressures are measured should be source documented.

If the subject is reporting symptoms of orthostatic hypotension when standing up after the blood pressure measurement, then the subject will be asked to lie down for 5 minutes, blood pressure and pulse rate will be measured, then the subject will be asked to stand and blood pressure and pulse rate measurements will be repeated after standing 1 to 3 minutes in order to measure the severity of the orthostatic hypotension. Vital signs will be collected at Baseline, at all visits from Week 2 through Week 52, and at unscheduled visits.

### 6.4.3 Electrocardiograms

All 12-lead ECGs will be complete, standardized recordings, performed in triplicate whenever possible at Baseline, and at all visits from Week 2 through Week 52 visits. The involvement of experienced personnel in the conduction of ECG recording in this population is strongly recommended.

Electrocardiograms should be performed before blood sampling or at least 30 minutes after blood sampling. The subject must rest in a sitting or supine position for 5 minutes before the ECG is obtained. Mild sedation is allowed exceptionally for ECGs (e.g., alprazolam at a pediatric-appropriate dose per age, and the *lowest dose* deemed necessary by the Investigator)


just in cases when the subject's agitation/anxiety does not allow a safe and accurate measurement and the Investigator, with agreement from the caregiver, considers it safe and appropriate for the subject. ECG tracings (paper or electronic) will be reviewed and interpreted by a qualified clinician. ECG tracings and results (ventricular rate, PR, QRS, QT, QTcF, and corrected QT interval using Bazett's correction method [QTcB] intervals) will be included in the subject's

Eligibility at Baseline should be based on ECG tracings collected on the study-provided ECG device during the visit and on the ECG central read. All ECGs will be centrally read; the cardiology central overread is considered final. The QTcF/QRS as well as other exclusionary values and abnormalities of all the tracings of adequate quality will be reviewed to determine eligibility.

A maximum of one repeat ECG procedure is allowed at Baseline.

### **6.4.4** Laboratory Evaluations

study records.

Clinical laboratory sample collection (including HbA<sub>1c</sub>) is encouraged, but not required, to be completed under fasting conditions. The laboratory evaluations will include, but are not limited to, the following:

- Clinical chemistry serum tests
  - Sodium (Na), potassium (K), carbon dioxide (CO<sub>2</sub>), chloride (Cl), phosphorus (P),
     calcium (Ca), blood urea nitrogen (BUN), creatinine (CR), glucose, albumin (ALB),
     total protein



- Alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), alkaline phosphatase (ALP), total bilirubin (TBIL), lactate dehydrogenase (LDH)
- Lipid panel


- Total cholesterol, high-density lipoprotein (HDL)-cholesterol, triglycerides, low-density lipoprotein (LDL)-cholesterol, cholesterol/HDL ratio, non-HDL cholesterol
- o HbA<sub>1c</sub>
- o Prolactin



- o Creatine kinase (CK)/creatine phosphokinase (CPK)
- Pregnancy test
  - A urine pregnancy test should be performed at all designated visits (Table 6–1) for women of child-bearing potential. If positive, the result will be confirmed with a serum pregnancy test.
    - If urine cannot be obtained in women of childbearing potential, a serum pregnancy test should be done in its place
- Hematology tests
  - o Complete blood count (CBC) including:
    - White blood cell (WBC) count
    - Complete differential (relative and absolute)
    - Hematocrit (Hct), hemoglobin, red blood cells (RBC), platelets
    - Reticulocyte count
- Urinalysis
  - o Blood, RBCs, WBCs, protein, glucose, ketones, specific gravity, pH
  - Reasonable efforts should be made to collect a urine sample from all subjects. When collection of a urine sample proves impractical or impossible (e.g., because the subject is incontinent or unable to cooperate), failure to collect a urine sample should be recorded in the subject's eCRF, and will not be considered a protocol deviation.
- Urine toxicology screen
  - O Urine toxicology screen will test for controlled substances. The following controlled substances may be tested with a urine toxicology screen according to the schedule presented in Table 6–1: amphetamine, barbiturates, benzodiazepines, cocaine, methadone, morphine/opiates, methamphetamine, marijuana (tetrahydrocannabinol [THC]), phencyclidine (PCP), ecstasy (3,4-methylenedioxymethamphetamine [MDMA]). A negative drug screen is required for study eligibility.


 Subjects who test positive and have a valid prescription for a controlled substance may be retested if they agree to abstain from the medication for the length of their participation in the study. The repeat test, and any other tests, must be negative for

them to participate in the study.

Laboratory evaluations will be completed according to the schedule presented in Table 6–1 and procedures detailed in the study laboratory manual. Additional safety testing may be performed at the discretion of the Investigator or designee.

Table 6–1 Safety Laboratory Evaluations

| Visit | Tests |
|---|---|
| Visit 1 (Baseline) | CHEM, CBC, UA, urine toxicology screen and dipstick, urine pregnancy test |
| Visit 2 (Week 2) | Urine pregnancy test |
| Visit 3 (Week 6) | Urine pregnancy test |
| Visit 4 (Week 12) | CHEM, CBC, UA, urine pregnancy test |
| Visit 5 (Week 20) | Urine pregnancy test |
| Visit 6 (Week 28) | CHEM, CBC, UA, urine pregnancy test |
| Visit 7 (Week 36) | Urine pregnancy test |
| Visit 8 (Week 44) | CHEM, CBC, UA, urine pregnancy test |
| Visit 9 (ET/EOT) | CHEM, CBC, UA, urine toxicology screen, urine pregnancy test |

Abbreviations: CBC=complete blood count; CHEM=clinical chemistry serum tests; EOT=end of treatment; ET=early termination; UA=urinalysis

### 6.4.5 Syncope

At each study visit, the investigator should query the caregiver for occurrences of syncope since the last visit. An occurrence of syncope should be reported as an adverse event. If the caregiver reports an occurrence of syncope, the investigator should ask the "syncope adverse event questions" in Appendix G.

### 6.4.6 Somnolence

At each study visit, the investigator should query the caregiver for occurrences of somnolence since the last visit. An occurrence of somnolence should be reported as an adverse event. If the caregiver reports an occurrence of somnolence, the investigator should ask the "somnolence adverse event" questions in Appendix H.


### 6.5 Blood Sampling

The involvement of experienced personnel in the conduction of blood drawing in this population is strongly recommended.

During blood sampling, measures to reduce pain are encouraged and can include application of numbing medication (e.g., lidocaine/prilocaine cream) to the draw site and/or use of a winged infusion set (i.e., a "butterfly" needle). Mild sedation is allowed exceptionally for blood draws (e.g., alprazolam at a pediatric-appropriate dose per age, and the *lowest dose* deemed necessary by the Investigator) just in cases when the subject's agitation/anxiety does not allow a safe and accurate measurement and the Investigator, with agreement from the caregiver, considers it safe and appropriate for the subject.

The total amount of blood to be obtained from each subject for safety laboratory blood samples during the course of this study will not exceed approximately 40 mL (6- through 17-year-olds) and 31.1 mL (5-year-olds). Note: this total amount does not account for additional blood samples that may be collected (e.g., to verify elevated laboratory results, etc.).

Table 6–2 tabulates the maximum allowable blood collection volumes by weight for affected children and Table 6–3 and Table 6–4 summarize the blood volumes to be drawn from 6-through 17-year-olds and 5-year-olds, respectively, in both a 24-hour and a 30-day period. The total amount of blood to be obtained from each subject should not exceed the allowable limits for affected children.

Table 6–2 Blood Collection Volume Limits in Affected Children

| Weight | 14 kg | 15 kg | 16 kg | 17 kg |
|---|---|---|---|---|
| Maximum allowable blood volume in a 24-hour period | 28 mL | 30 mL | 32 mL | 34 mL |
| Maximum allowable blood volume in a 30-day period | 56 mL | 60 mL | 64 mL | 68 mL |

Sources: North Shore LIJ Human Subject Protection Program Guidance Document, Maximum Blood Draw Limits, Version 11/24/14; National Center for Health Statistics (CDC) 2-20 years: Stature-for-age and weight-for-age percentiles

Notes: 5th percentile body weight for 5 year old girls≈14.6 kg; 5th percentile body weight for 5 year old boys≈15.1 kg.


Table 6–3 Blood Collection Volumes for Safety Labs (6- through 17-year-olds)

| | Baseline<br>Visit | Visit 4<br>(Week 12) | Visit 6<br>(Week 28) | Visit 8<br>(Week 44) | Visit 9<br>(Week 52) |
|---|---|---|---|---|---|
| Total safety labs each study visit | 8 mL | 8 mL | 8 mL | 8 mL | 8 mL |
| Total volume in any 24-hour period | 8 mL | 8 mL | 8 mL | 8 mL | 8 mL |
| Total volume in any 30-day period | | | | | |
| Baseline | 8 mL | | | | |
| Week 12 | | 8 mL | | | |
| Week 28 | | | 8 mL | | |
| Week 44 | | | | 8 mL | |
| Week 52 | | | | | 8 mL |

Table 6-4 Blood Collection Volumes for Safety Labs (5-year-olds)

| | Baseline<br>Visit | Visit 4<br>(Week 12) | Visit 6<br>(Week 28) | Visit 8<br>(Week 44) | Visit 9<br>(Week 52) |
|---|---|---|---|---|---|
| Total safety labs each study visit | 5.9 mL | 6.3 mL | 6.3 mL | 6.3 mL | 6.3 mL |
| Total volume in any 24-hour period | 5.9 mL | 6.3 mL | 6.3 mL | 6.3 mL | 6.3 mL |
| Total volume in any 30-day period | | | | | |
| Baseline | 5.9 mL | | | | |
| Week 12 | | 6.3 mL | | | |
| Week 28 | | | 6.3 mL | | |
| Week 44 | | | | 6.3 mL | |
| Week 52 | | | | | 6.3 mL |

### 6.6 Safety Follow-up

A 30-day safety follow-up telephone contact is to be completed for subjects who complete the treatment period of the study, as well as those who discontinue prematurely from the study. Subjects should have the following completed at 30(+3) days after last dose of study drug:

- Assessment of concomitant medications/treatments
- Assessment of AEs
- Assessment of syncope

• Assessment of somnolence

### 6.7 Unscheduled Visits

Unscheduled visits may occur as determined by the Investigator. The following safety assessments generally should be recorded at each unscheduled visit: assessment of AEs, assessment of syncope, assessment of somnolence, assessment of concomitant medications/treatments, measurement of vital signs and weight, the ESRS-A, and completion of the C-SSRS. The Investigator may perform any additional safety evaluations deemed by the Investigator to be clinically indicated.

### **6.8** Remote Assessments or Visits

Circumstances may arise (e.g., pandemic, natural disaster, political upheaval, or to minimize subject and caregiver burden) when on-site assessments of efficacy and/or safety are not possible. In those cases, assessments may be performed offsite by raters either in person, or via video technology or telephone where possible. For all visits that are conducted remotely, the Investigator <u>must</u> contact the Medical Monitor for approval of the plan. Sites must keep a log to identify details of all visits that are administered remotely. For some remote efficacy assessments the vendor will provide additional training to ensure calibration to reduce discrepancy between on-site and remote assessments (ABC, CGI-S, RBS-R, VABS-Socialization).

Provided that the subject is physically in the clinic, and accompanied by a relative, all caregiver-rated assessments may be provided remotely.

### 7 ADVERSE EVENTS

### 7.1 Specification of Safety Parameters

### 7.1.1 Definition of Adverse Event

An AE is defined as "any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study drug, whether or not considered related to study drug".

An AE can therefore be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality or seriousness. An AE can arise from any use of the drug (e.g., off-label use, use in combination with another drug) and from any route of administration, formulation, or dose, including an overdose.

A suspected adverse reaction is any AE for which there is a reasonable possibility that the drug caused the AE.


Study: ACP-103-070 Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

AEs do not include the following:

• Stable or intermittent chronic conditions (such as myopia requiring eyeglasses) that are present prior to Baseline and do not worsen during the study

- Medical or surgical procedures (e.g., surgery, endoscopy, tooth extraction, transfusion), or scheduled surgery/procedure. The condition that leads to the procedure is an AE if not present at time of consent.
- Overdose of <u>concomitant</u> medication without any signs or symptoms will not be considered an AE, but if a subject is hospitalized or has other serious criteria, the overdose will be considered an AE and shall be reported on the Sponsor's Overdose Reporting form.
- Hospitalization for elective surgery planned prior to study (situation where an untoward medical occurrence has not occurred)
- Pregnancy will not be considered an AE, but if it occurs, it will be reported on a pregnancy form

### 7.1.2 Definition of Serious Adverse Event

In addition to the severity rating, each AE will be classified by the Investigator as "serious" or "not serious." The seriousness of an event will be defined according to the applicable regulations and generally refers to the outcome of an event. An SAE is one that meets one or more of the following:

- Is fatal
- Is life threatening
- Results in disability or permanent damage
- Requires hospitalization (initial or prolonged)
- Results in congenital anomaly or birth defect
- Other serious event (medically significant/important medical event)

### **Definition of Life Threatening**

A life threatening event places the subject at <u>immediate</u> risk of death from the event as it occurred. This does not include an AE, which, had it occurred in a more severe form, might have caused death.

### **Definition of Hospitalization**

Hospitalization is defined by the Sponsor as a full admission to the hospital for diagnosis and treatment. This includes prolongation of an existing inpatient hospitalization.

Study: ACP-103-070 Clinical Study Protocol Amendment 3-Consolidated

Clinical Study Protocol Amendment 3-Consolidated

Date: 29 February 2024

Examples of visits to a hospital facility that do **not** meet the serious criteria for hospitalization

• Emergency room visits (that do not result in a full hospital admission)

Outpatient surgery

include:

- Preplanned or elective procedures
- Protocol procedures
- Social hospitalization, defined as admission to the hospital as a result of inadequate family support or care at the subject's primary residence

### **Definition of Disability or Permanent Damage**

Disability is defined as a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.

### **Definition of Medically Significant**

Important medical events (medically significant events) that may not result in death, be life threatening, or require hospitalization may be considered to be an SAE when, based upon appropriate medical judgment, they may jeopardize the subject or may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

An SAE may also include any other event that the Investigator or Medical Monitor judges to be serious or that suggests a significant hazard, contraindication, side effect, or precaution.

### 7.2 Classification of an Adverse Event

### 7.2.1 Severity of Event

The severity of each AE will be assessed as described below and reported in detail as indicated on the eCRF:

- Mild: awareness of sign or symptom but easily tolerated, causing minimal discomfort, and not interfering with normal everyday activities
- Moderate: sufficiently discomforting to interfere with normal everyday activities
- Severe: incapacitating and/or preventing normal everyday activities

### 7.2.2 Relationship to Study Drug

The causality of each AE should be assessed and classified by the Investigator as "related" or "not related." An event is considered related if there is a reasonable possibility that the event may


have been caused by the product under investigation (i.e., there are facts, evidence, or arguments to suggest possible causation).

### Consider the following when assessing causality:

- Temporal associations between the agent and the event
- Response to drug cessation (de-challenge) or re-challenge
- Compatibility with known class effect
- Known effects of concomitant medications
- Pre-existing risk factors
- A plausible mechanism
- Concurrent illnesses
- Past medical history

### 7.2.3 Duration

The start and stop dates for AEs will be recorded using the following criteria:

- Start: Date of the first episode of the AE or date of worsening in severity
- Stop: Date when AE recovered or resolved, recovered or resolved with sequelae, or worsened in severity

### 7.2.4 Frequency

The frequency of the AE should be indicated according to the following definitions:

- Single: Experienced once, without recurrence at same severity
- **Recurrent:** More than one discrete episode with the same severity

### 7.2.5 Action Taken With Study Drug

- **Dose not changed:** No change in study drug
- **Dose increased:** Study drug dose increased (can only be done up to and including Week 20 visit)
- **Dose reduced:** Study drug dose reduced (can only be done up to and including Week 20 visit)
- Drug interrupted: Study drug temporarily stopped
- Drug withdrawn: Study drug discontinued permanently
- Not applicable
- Unknown


Study: ACP-103-070 Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

### 7.2.6 Therapy

• None: No new treatment instituted

Medication: New treatment initiated as a direct result of AE

• Other: Other action required

### **7.2.7 Outcome**

Recovered/resolved: Recovered or resolved

• Recovered/resolved with sequelae: Recovered or resolved with sequelae

Not recovered/not resolved: Not recovered or not resolved

• **Fatal:** Death due to an AE

Unknown: Unknown

### 7.2.8 Seriousness

Not serious

• Serious (see Section 7.1.2)

### 7.2.9 Definition of Unexpectedness

An AE, the nature or severity of which is not consistent with the information provided in the Reference Safety Information section of the current pimavanserin Investigator's Brochure.

### 7.3 Time Period and Frequency for Event Assessment and Follow-up

Adverse events will be recorded from the first dose of open-label study drug through the study safety follow-up period. All ongoing AEs from the antecedent double-blind study will be carried over and recorded from Baseline for the ACP-103-070 study until resolution or the follow-up safety assessment. If an AE is ongoing at the end of the study safety follow-up period, every reasonable attempt should be made to follow and appropriately treat the subject until the AE resolves or until the Investigator deems the AE to be chronic or stable.

In the event that a subject discontinues from the study and has an ongoing AE at the time of discontinuation (Section 4.5.1), the subject should be followed and appropriately treated until the AE resolves or until the Investigator deems the AE to be chronic or stable. If a subject withdraws from the study because of an AE, no additional assessments may be performed (Section 4.4).

### 7.4 Reporting Procedures

### 7.4.1 Adverse Event Reporting

The Investigator must record all observed AEs and all reported AEs. At each visit, the Investigator should ask the subject a nonspecific question (e.g., "Have you noticed anything

Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

different since your last visit?") to assess whether any AEs have been experienced since the last report or visit.

Note that any use of medication (and specifically any newly prescribed medication) during the course of a study may indicate the occurrence of an AE that may need to be recorded on both the AE and the concomitant medication page.

All AEs, serious and not serious, will be recorded on the AE eCRF page using appropriate medical terminology. Severity and relationship to study drug will be assessed by the Investigator.

When possible, clinical AEs should be described by diagnosis and not by symptoms (e.g., "cold" or "seasonal allergies" instead of "runny nose").

All AEs, whether or not related to the study drug, must be fully and completely documented on the AE eCRF and in the subject's notes.

### 7.4.2 Serious Adverse Event Reporting

The reporting of SAEs by the Sponsor or designee to the regulatory authorities is a regulatory requirement. Each regulatory authority has established a timetable for reporting SAEs based upon established criteria.

Serious AEs must be reported within 24 hours of discovery to the Sponsor or its designee; both using the appropriate form for initial and/or follow-up reporting and entering in the electronic data capture (EDC) system.

At a minimum, events identified by the Sponsor to require expedited reporting as serious, unexpected, and related to study drug must be brought to the attention of the responsible IRB/EC, as per applicable regulations. These will be provided by the Sponsor after their assessment. For European Union member states, the Sponsor or its designee will provide reports of suspected unexpected serious adverse reactions (SUSARs) directly to the ECs, as required by local legislation. In all other countries, it is the Investigator's responsibility to provide these expedited reports to the responsible IRB/EC. It is also the Investigator's responsibility to notify the responsible IRB/EC regarding any new and significant safety information.

When an SAE occurs, Investigators will review all documentation related to the event and will complete the paper SAE form, as well as enter the SAE into the EDC system, with all required information (for initial and/or follow-up information) and fax or email (within 24 hours of discovery) to the contact information provided on the SAE form.

Subjects will be followed through the safety follow-up period (i.e., 30[+3] days after last dose of study drug) for any SAEs and/or other reportable information until such events have resolved or the Investigator deems them to be chronic or stable.


feasible following the report of the SAE.

In the event of any SAE (other than death), the study subject will be instructed to contact the Investigator (or designee) using the telephone number provided in the informed consent form (ICF). All subjects experiencing an SAE will be seen by the Investigator or designee as soon as is

Serious AEs occurring after the safety follow-up period (i.e., 30[+3] days after last dose of study drug) should be reported if in the judgment of the Investigator there is "a reasonable possibility" that the event may have been caused by the product.

SAEs should also be reported to the IRB/EC according to local regulations.

### 7.4.3 Reporting of Pregnancy

Any female subject who becomes pregnant during the study (with or without AEs) must be discontinued from the study and the pregnancy must be reported on the Pregnancy form within 24 hours of discovery to the Sponsor or its designee. Any female subject who becomes pregnant during the study will be followed through the pregnancy outcome.

Any AEs that are the consequence of pregnancy and which meet the criteria for serious should also be reported via the SAE form.

### 7.4.3.1 Reporting Paternal Drug Exposure

Paternal drug exposure is defined as a father's exposure to a medicinal product before or during his partner's pregnancy. Any paternal drug exposure cases must be reported to the Sponsor within 24 hours of discovery via the Pregnancy form. Any AEs that are the consequence of paternal drug exposure and which meet the criteria for serious must also be reported to the Sponsor within 24 hours of discovery via the SAE form.

### 7.4.4 Reporting of Overdose

An overdose is a deliberate or inadvertent administration of a treatment at a dose higher than the maximum recommended dose per protocol. It must be reported to the Sponsor or designee on the Sponsor Overdose Reporting form within 24 hours of discovery. In addition, all events of overdose are to be captured as protocol deviations (see Section 5.1.6).

### 8 MONITORING

Routine monitoring of study sites is described in Section 11.

Clinical site monitoring is conducted to ensure that the rights and well-being of human subjects are protected, that the reported study data are accurate, complete, and verifiable, and that the conduct of the study is in compliance with the currently approved protocol and amendment(s) as applicable, with GCP, and with applicable regulatory requirements. Details of the study site monitoring process are described in a separate clinical monitoring plan document.


### 9 STATISTICAL METHODS AND DATA ANALYSIS

### 9.1 Statistical and Analytical Plans

Statistical methods will be documented in detail in a statistical analysis plan (SAP) to be approved by the Sponsor prior to database lock. Deviations from the approved SAP, if any, will be described and justified in the final clinical study report.

### 9.2 Statistical Hypotheses

The primary objective of this study is to evaluate the long-term safety and tolerability of pimavanserin after 52 weeks of treatment in children and adolescents with ASD. Secondary and exploratory objectives include assessment of efficacy outcome measures over time. No formal statistical testing will be performed for any of the safety or efficacy endpoints.

All safety and efficacy measures will be summarized descriptively.

### 9.3 Sample Size Determination

The planned sample size for this study is not based on statistical power but will depend on the number of subjects who complete the antecedent double-blind study, and who rollover into this open-label extension study.

Assuming a drop-out rate of 15% in the antecedent study, it is estimated that approximately 193 subjects will be eligible to enroll in this OLE. Assuming all 193 subjects do enroll, then according to the Rule of Three, the 95% confidence interval for the occurrence rate of an unobserved adverse event is estimated as (0, 1.6%).

### 9.4 Population Analysis Sets

The **Safety Analysis Set** will include all subjects who received at least one dose of open-label study drug. The Safety Analysis Set will be used for all analyses.

### 9.5 Statistical Analyses

For continuous variables, the following summary statistics will be provided: number of subjects, mean, standard error of the mean, standard deviation, minimum, maximum, and median. For categorical variables, summaries will include the number and percentage of subjects in each category.

For each continuous measure in safety and efficacy analyses, changes from Baseline results will be presented in two ways:

1. using the Baseline of this study to report the changes across the timepoints of this open-label study


the timepoints of this open-label study

2. using the Baseline from the antecedent double-blind study to report the changes across

### 9.5.1 Primary Analyses

The primary endpoints for this study are TEAEs. All adverse events will be classified into standard terminology using the Medical Dictionary for Regulatory Activities (MedDRA). A TEAE is defined as an AE that started after first study dose administration and no later than last study dose date +30 days. The number and frequency of TEAEs will be summarized by system organ class and preferred term. TEAEs leading to discontinuation, TEAEs related to study drug, TEAEs by maximum severity, fatal TEAEs, serious TEAEs, and serious TEAEs related to study drug will also be summarized.

### 9.5.2 Other Safety Analyses

Descriptive summary statistics for ECGs, vital signs, weight, BMI, ESRS-A, and clinical laboratory parameters, including changes from Baseline, will be tabulated by timepoint. Additionally, categorical analyses will be conducted on the incidence of subjects with prolonged QTc intervals and changes in QTc intervals in accordance with ICH guidelines.

For the C-SSRS, the number and percentage of subjects with suicidal ideation or behavior during the study will be tabulated.

### 9.5.3 Secondary Endpoint and Analysis

The secondary endpoint in this study is the proportion of subjects who have at least 25% reduction from the antecedent study Baseline in the ABC-Irritability (ABC-I) subscale score AND a CGI-I of irritability score of 1 (very much improved) or 2 (much improved) compared to the antecedent study baseline status at Week 52.

The number and percentage of subjects who have at least 25% reduction from antecedent-study Baseline in the ABC Irritability (ABC-I) subscale score AND a CGI-I of irritability score of 1 (very much improved) or 2 (much improved) compared to the antecedent study baseline status will be tabulated by timepoint.

### 9.5.4 Exploratory Endpoints and Analyses

Exploratory endpoints are the following:

- Change from Baseline at Week 52 in the caregiver-rated ABC subscale scores
  - Irritability
  - o Stereotypic behavior
  - Lethargy
  - Hyperactivity


Study: ACP-103-070
Clinical Study Protocol Amendment 3-Consolidated

Inappropriate speech

- Change from Baseline at Week 52 in the CGI-S of irritability score
- CGI-I of irritability score compared to the antecedent study baseline status at Week 52
- Change from Baseline at Week 52 in the CGSQ scores
- Proportion of subjects who have at least 25% reduction from the antecedent study Baseline in the ABC-I subscale score (ABC-I responders) at Week 52
- Proportion of subjects who have CGI-I of irritability score of 1 (very much improved) or 2 (much improved) compared to the antecedent study baseline status (CGI-I of irritability responders) at Week 52

Descriptive summary statistics for each of the ABC subscale score, CGI-S of irritability score, CGI-I of irritability score and CGSQ score, and associated change from Baseline values (except for CGI-I of irritability), will be tabulated by timepoint.

The number and percentage of subjects who have at least 25% reduction from Baseline in the ABC-I subscale score, and the number and percentage of subjects with CGI-I of irritability score of 1 (very much improved) or 2 (much improved) compared to the antecedent-study baseline status will also be tabulated by timepoint.

### 9.5.5 Subgroup Analyses

Selected analyses may be performed in subgroups defined in the SAP.

### 9.6 Interim Analyses

No interim analyses are planned for this study.

### 9.7 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review interim safety data, including data on AEs, SAEs and safety laboratory data. The DSMB will be independent of the Sponsor and the Investigators and will be empowered to recommend stopping the study due to safety concerns. The membership, activities, responsibilities, and frequency of meetings will be described separately in the DSMB charter.

### 10 STUDY MANAGEMENT AND DATA COLLECTION

### 10.1 Data Collection and Management Responsibilities

All documents required for the conduct of the study as specified in the ICH GCP guidelines will be maintained by the Investigator in an orderly manner and made available for monitoring and/or auditing by the Sponsor and regulatory authorities.

The Investigator and institution must permit authorized representatives of the Sponsor or designees (including monitors and auditors), regulatory authorities (including inspectors), and the IRB/EC direct access to source documents (such as original medical records) as allowed by local regulations. Direct access includes permission to examine, analyze, verify, and reproduce any records and reports that are needed for the evaluation of the study either in person or through remote video/electronic medium (such as email) if applicable. The Investigator must ensure the reliability and availability of source documents from which the information on the eCRF was derived.

## 10.2 Source Documents

All study specific information obtained at each study visit must be recorded in the subject's record (source documentation), and then entered into a validated EDC database by trained site personnel. The source documentation may consist of source notes captured by site personnel in laboratory reports, ECG reports, and electronic source data.

## **10.3** Case Report Forms

Subject data required by this protocol are to be recorded in an EDC system on eCRFs and/or captured electronically by data vendors. The Investigator and his or her site personnel will be responsible for completing the eCRFs. The Investigator is responsible for the accuracy and reliability of all the information recorded on the eCRFs. All information requested on the eCRFs needs to be supplied, including subject identification data, visit date(s), assessment values, etc., and any omission or discrepancy will require explanation. All information on eCRFs must be traceable to source documentation (unless eCRF is considered the source) at the site.

## **10.4** Confidentiality

The Investigator must ensure that each subject's anonymity is maintained as described below. On the eCRFs, medical records, or other documents submitted to the Sponsor or designees, subjects must be identified by a subject identification number only. Subject identifiers uniquely identify subjects within the study and do not identify any person specifically. Documents that are not for submission to the Sponsor or designees (e.g., signed ICFs) should be kept in strict confidence by the Investigator in compliance with Federal regulations or other applicable laws or ICH guidance on GCP. Data collection and handling should comply with the European Union General Data Protection Regulation (EU GDPR) and other relevant regulations concerning data privacy, where applicable. Acadia has assigned a Data Protection Officer (DPO) as per the EU GDPR.

## 10.5 Study Records Retention

Investigators are required to maintain all essential study documentation as per ICH GCP guidelines. This includes, but is not limited to, copies of signed, dated and completed


eCRFs, documentation of eCRF corrections, signed ICFs, audio recordings, subject-related source documentation, and adequate records for the receipt and disposition of all study drug. Investigators should maintain all essential study documentation, for a period of at least 2 years following the last approval of marketing application in an ICH region (US, Europe, and Japan), or until at least 2 years after the drug investigational program is discontinued, unless a longer period is required by applicable law or regulation. Only the Sponsor can notify an Investigator or vendor when any records may be discarded. Investigators should contact the Sponsor before

## 10.6 Protocol Exceptions and Deviations

destroying any files.

No prospective entry criteria protocol deviations are allowed; all subjects must meet all eligibility criteria in order to participate in the study.

Protocol waivers for eligibility will not be granted by the Sponsor under any circumstances. If, during the course of a subject's post-enrollment participation in the trial it is discovered that the subject did not meet all eligibility criteria, this will be reported as a major protocol deviation and not a waiver. In this situation, the subject will be discontinued, unless the discontinuation presents an unacceptable medical risk. The justification to allow the subject to continue in the trial will be made by the Sponsor, with medical input from the Investigator, and will be documented. All follow-up safety assessments must be completed and documented as outlined in the protocol (Section 6.6). The Investigator must report any protocol deviation to the Sponsor and, if required, to the IRB/EC in accordance with local regulations, within reasonable time.

#### 10.7 Protocol Amendments

Changes to the protocol may be made only by the Sponsor (with or without consultation with the Investigator). All protocol modifications must be submitted to the site IRB/EC in accordance with local requirements and, if required, to regulatory authorities, as either an amendment or a notification. Approval for amendments must be awaited before any changes can be implemented, except for changes necessary to eliminate an immediate hazard to trial subjects, or when the changes involve only logistical or administrative aspects of the trial. No approval is required for notifications.

## 11 QUALITY MANAGEMENT

## 11.1 Risk Management

The Sponsor utilizes the ICH E6 (GCP) Revision 2 risk management approach that includes methods to assure and control the quality of the trial proportionate to the risks inherent in the trial and the importance of the information collected. The intent is that all aspects of this trial are


operationally feasible and that any unnecessary complexity, procedures, and data collection are avoided. The Sponsor's risk management approach includes the following documented activities:

- Critical Process and Data Identification: during protocol development, risks of processes and data that are critical to ensure human subject protection and the reliability of trial results are identified and assessed.
- Risk Identification: risks to critical trial processes, governing systems, investigational product, trial design, data collection, and recording are identified.
- Risk Evaluation: identified risks are evaluated by considering the following factors: (a) likelihood of occurrence, (b) impact on human subject protection and data integrity, and (c) detectability of errors.
- Risk Control: risks that can be avoided, reduced (i.e., mitigated), or accepted are differentiated. Risk mitigation activities are incorporated in protocol design and implementation, study plans, training, processes, and other documents governing the oversight and execution of study activities. Where possible, predefined quality tolerance limits are defined to identify systematic issues that can impact subject safety or data integrity and deviations from the predefined quality tolerance limits will trigger an evaluation and possibly an action. Contingency plans are developed for issues with a high risk factor that cannot be avoided.
- Periodic risk review, communication, and escalation of risk management activities during trial execution and risk outcome reporting in the clinical study report (CSR).

### 11.2 Quality Control and Quality Assurance

The Sponsor or designees and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., eCRFs and other pertinent data) provided that subject confidentiality is respected.

The Sponsor's or designee's monitor is responsible for inspecting the eCRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to subject medical records and other study-related records needed to verify the entries on the eCRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits are resolved.

In accordance with ICH guidance on GCP and the Sponsor's audit plans, sites participating in this study may be audited. These audits may include a review of site facilities (e.g., pharmacy, Clinical Study Protocol Amendment 3-Consolidated

Date: 29 February 2024

drug storage areas, and laboratories) and review of study-related records may occur in order to
evaluate the trial conduct and compliance with the protocol, ICH guidance on GCP, and

The Sponsor's or designee's representatives, regulatory authority inspectors and IRB/EC representatives who obtain direct access to source documents should also respect subject confidentiality, taking all reasonable precautions in accordance with applicable regulatory requirements to maintain the confidentiality of subjects' identities.

## 12 ETHICAL CONSIDERATIONS

applicable regulatory requirements.

#### 12.1 Ethical Standard

The study will be conducted in compliance with the protocol, the Declaration of Helsinki, ICH GCP, and other applicable regulatory requirements (e.g., Serious Breach reporting, urgent safety measures, and European Union General Data Protection Regulation [EU GDPR]).

The study will be performed in accordance with current US Health Insurance Portability and Accountability Act (HIPAA) regulations, US FDA GCP Regulations (US CFR 21 parts 50, 54, 56, and 312), and ICH guidance on GCP (E6) and clinical safety data management (E2A).

In accordance with Directive 75/318/EEC, as amended by Directive 91/507/EEC, the final clinical study report will be signed by an Investigator and/or Coordinating Investigator who will be designated prior to the writing of the clinical study report.

## 12.2 Institutional Review Board/Ethics Committee

The Investigator or designee will provide the IRB/EC with all requisite material, including a copy of the protocol, informed consent, any subject information or advertising materials, and any other requested information. The study will not be initiated until the IRB/EC provides written approval of the protocol and the informed consent and until approved documents have been obtained by the Investigator and copies received by the Sponsor. All amendments will be sent to the IRB/EC for information (minor amendment) or for submission (major amendment) before implementation. The Investigator will supply the IRB/EC and the Sponsor with appropriate reports on the progress of this study, including any necessary safety updates, in accordance with the applicable government regulations and in agreement with policy established by the Sponsor.

## 12.3 Informed Consent/Assent Process

Properly executed, written informed assent/consent must be obtained from each subject and/or subject's parent/LAR prior to any Baseline procedures.

The informed consent must, at a minimum, include the elements of consent described in the ICH guidance on GCP and the US CFR 21 part 50.25. A copy of the ICF planned for use will be


reviewed by the Sponsor or designee for acceptability and must be submitted by the Investigator or designee together with the protocol, to the appropriate IRB/EC for review and approval prior to the start of the study at that investigational site. Consent forms must be in a language fully comprehensible to the prospective subject and their parent/ LAR. The Investigator must provide the Sponsor or designee with a copy of the IRB/EC letter approving the protocol and the ICF before the study drug supplies will be shipped and the study can be initiated.

The consent form must be revised if new information becomes available during the study that may be relevant to the subject's willingness to continue participation. Any revision must be submitted to the appropriate IRB/EC for review and approval in advance of use.

## 12.3.1 Subject Assent Form

To participate in the study, the subject will assent to an understanding of, and sign the assent form. The subject will be made aware of the ability to withdraw from the study at any time, without prejudice. The subject's assent for participation must be documented. Assent is the affirmative agreement to participate in the research of a minor. If the subject cannot sign the form, a witness will be allowed to provide written verification of oral assent

## 12.3.2 Parent and Legally Acceptable Representative Informed Consent

Written informed consent will be obtained from the subject's parent/LAR before the subject participates in any study-related procedure. To provide consent for the subject's participation in the study, the subject's parent/LAR will read, assent to an understanding of, and sign an ICF or other locally applicable regulations and authorization form after having had an opportunity to discuss the forms with the Investigator. The parent/LAR will be made aware that the subject may withdraw from the study at any time and will receive a copy of the signed ICF. Subjects who reach the age of majority (i.e., 18 years in most jurisdictions) during the course of the study are required to be re-consented.

### 12.3.3 Consent and Other Informational Documents Provided to Subjects

The subject and/or parent/LAR must be given a copy of the signed informed consent and the original maintained in the designated location at the site.

#### 12.3.4 Consent Procedures and Documentation

It is the Investigator or designee's responsibility to obtain written informed consent from the subject and/or parent/LAR after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study. The subject and/or parent/LAR must be given ample time to decide about study participation and opportunity to inquire about details of the study. The IRB/EC-approved consent form must be personally signed and dated by the subject or parent/LAR with subject assent and by the person who conducted the informed-consent discussion. The


in the subject's study documents.

Investigator or appropriate site personnel must document the details of obtaining informed consent

Records related to a study subject's participation will be maintained and processed according to local laws, and where applicable, the European Union General Data Protection Regulation (EU GDPR). The consent and study information documentation will include statements describing local and regional requirements concerning data privacy, and who to contact for questions.

#### 12.3.4.1 Remote Consent Procedures and Documentation

In exceptional circumstances, and with the approval of the Medical Monitor, Investigators may obtain informed consent from the subject or parent/LAR when these individuals are unable to travel to the site where the Investigator is located due to extenuating circumstances (e.g., pandemic, natural disaster, or political upheaval). This is only permitted when a new consent is approved by the IRB/EC and the subject and/or parent/LAR need to be re-consented. The consent form may be sent to the subject or the subject's parent/LAR by facsimile or e-mail, and the consent interview may then be conducted by telephone when the subject or subject's parent/LAR can read the consent form during the discussion. After the consent discussion, the subject or the subject's caregiver can sign and date the consent form. Options for returning the document to the clinical Investigator may include facsimile, scanning the consent form and returning it through a secure e-mail account, or posting it to a secure internet address. Alternatively, the subject or caregiver may bring the signed and dated consent form to his/her next visit to the clinical site, if restrictions on traveling to the clinical trial site are alleviated, or mail it to the clinical Investigator. The case history for each subject must document that informed consent was obtained prior to conducting any assessments at the visit the re-consent was conducted. The Investigator should have the subject and/or parent/LAR confirm verbally during the consent interview that the subject and/or parent/LAR has signed and dated the form. In addition, the person signing the consent form must receive a copy of the consent form.

### 13 PUBLICATION PLAN

All publication rights are delineated in the Clinical Study Agreement and/or other separate agreements with the Investigator and/or Institution, as applicable.

#### 14 CONFLICT OF INTEREST POLICY

## 14.1 Finance, Insurance, and Indemnity

Arrangements for finance, insurance, and indemnity are delineated in the Clinical Study Agreement and/or other separate agreements with the Investigator and/or Institution, as applicable.


#### 15 LITERATURE REFERENCES

Aaron E, Montgomery A, Ren X, et al. Whole blood serotonin and platelet 5-HT<sub>2A</sub> binding in autism spectrum disorder. *J Autism Dev Disord*. 2019;49(6):2417-2425.

Acadia Pharmaceuticals Inc. NUPLAZID® [package insert]. San Diego, CA, November 2020.

Akhondzadeh S, Erfani S, Mohammadi MR, et al. Cyproheptadine in the treatment of autistic disorder: a double-blind placebo-controlled trial. *J Clin Pharm Ther*. 2004;29(2):145-150.

Aldinger KA, Lane CJ, Veenstra-VanderWeele J, Levitt P. Patterns of risk for multiple co-occurring medical conditions replicate across distinct cohorts of children with autism spectrum disorder. *Autism Res.* 2015;8(6):771-781.

Aman MG, Singh NN, Stewart AW, Field CJ. Psychometric characteristics of the Aberrant Behavior Checklist. *Am J Ment Defic*. 1985;89(5):492-502.

Brannan AM, Heflinger CA, Bickman L. The Caregiver Strain Questionnaire: measuring the impact on the family of living with a child with serious emotional disturbance. *J Emot Behav Disord*. 1997;5(4):212-222.

Chouinard G, Margolese HC. Manual for the Extrapyramidal Symptom Rating Scale (ESRS). *Schizophr Res.* 2005;76(2-3):247-265.

Daly E, Ecker C, Hallahan B, et al. Response inhibition and serotonin in autism: a functional MRI study using acute tryptophan depletion. *Brain*. 2014;137(Pt 9):2600-2610.

Fung LK, Mahajan R, Nozzolillo A, Bernal P, Krasner A, Jo B, et al. Pharmacologic treatment of severe irritability and problem behaviors in autism: A systematic review and meta-analysis. *Pediatrics*. 2016;137(Suppl 2):S124-S135.

Grzadzinski R, Huerta M, Lord C. DSM-5 and autism spectrum disorders (ASDs): an opportunity for identifying ASD subtypes. *Mol Autism*. 2013;4:12.

Guy W. Clinical Global Impressions. In: ECDEU Assessment Manual for Psychopharmacology—Revised (DHEW publication number ADM 76–338). Rockville, MD, U.S. Department of Health, Education, and Welfare, Public Health Service, Alcohol, Drug Abuse, and Mental Health Administration, NIMH Psychopharmacology Research Branch, Division of Extramural Research Programs, 1976, 218-222.

Kaat AJ, Lecavalier L, Aman MG. Validity of the Aberrant Behavior Checklist in children with autism spectrum disorder. *J Autism Dev Disord*. 2014;44(5):1103-1116.

Lam KSL, Aman MG. The Repetitive Behavior Scale-Revised: independent validation in individuals with autism spectrum disorders. *J Autism Dev Disord*. 2007:37(5):855-866.


Levy SE, Mandell DS, Schultz RT: Autism. Lancet. 2009;374(9701):1627-1638.

Marshall WA, Tanner JM. Variations in the pattern of pubertal changes in girls. Arch Dis Child. 1969;44(235):291-303.

Marshall WA, Tanner JM. Variations in the pattern of pubertal changes in boys. Arch Dis Child. 1970;45(239):13-23.

McPheeters ML, Warren Z, Sathe N, et al. A systematic review of medical treatments for children with autism spectrum disorders. *Pediatrics*. 2011;127(5):e1312-e1321.

Muller CL, Anacker AM, Veenstra-VanderWeele J. The serotonin system in autism spectrum disorder: from biomarker to animal models. *Neuroscience*. 2016;321:24-41.

Paclt I, Hellerová P. [Ritanserin in autistic children]. Cesk Psychiatr. 1993;89(2):85-86.

Posner K, Brown GK, Stanley B, et al. The Columbia–Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. *Am J Psychiatry*. 2011;168(12):1266-1277.

Ritvo E, Yuwiler A, Geller E, Ornitz EM, Saeger K, Plotkin S. Increased blood serotonin and platelets in early infantile autism. *Arch Gen Psychiatry*. 1970;23(6):566-572.

Rolf L, Haarmann F, Grotemeyer K, Kehrer H. Serotonin and amino acid content in platelets of autistic children. *Acta Psychiatr Scand*. 1993;87:312-316.

Schwartz GJ, Muñoz A, Schneider MF, et al. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009;20:629-637.

Sharma SR, Gonda X, Tarazi FI. Autism spectrum disorder: classification, diagnosis and therapy. *Pharmacol Ther*. 2018;190:91-104.

Sparrow SS, Cicchetti DV, Saulnier CA. Vineland Adaptive Behavior Scales, Third Edition: Vineland-3. Pearson; 2016.

Vanover KE, Weiner DM, Makhay M, et al. Pharmacological and behavioral profile of N-(4-fluorophenylmethyl)-N-(1-methylpiperidin-4-yl)-N'-(4-(2-methylpropyloxy)phenylmethyl) carbamide (2R,3R)-dihydroxybutanedioate (2:1) (ACP-103), a novel 5-hydroxytryptamine(2A) receptor inverse agonist. *J Pharmacol Exp Ther.* 2006;317(2):910-918.


Study: ACP-103-070
Clinical Study Protocol Amendment 3-Consolidated

#### 16 APPENDICES

## Appendix A Prohibited and Restricted Medications<sup>a</sup>

Subjects taking prohibited medications at study entry will not be eligible for the study.

Subjects who require current treatment with a prohibited medication will be withdrawn from the study.

Subjects who have previously taken a prohibited medication during the study will be withdrawn from the study unless:

- the prohibited medication has been discontinued AND
- withdrawal from the study presents an unacceptable medical risk to the subject

The justification to allow the subject to continue in the trial will be made by the Sponsor/Medical Monitor with medical input from the Investigator, and will be documented. If allowed to remain in the trial, this will be reported as a major protocol deviation and not a waiver.

The table below lists prohibitions and restrictions by medication class, including representative medications within class. A **prohibited** medication is not allowed. A **restricted** medication is allowed only under certain conditions.

| <b>Medication Class</b> | Medicationa | Prohibition/restrictions |
|---|---|---|
| Antiarrhythmic | PROHIBITED | Prohibited at antecedent study entry and throughout the |
| drugs | • ajmaline | treatment period |
| | • amakalant, semantilide | |
| | • amiodarone | |
| | • bretylium | |
| | <ul> <li>disopyramide</li> </ul> | |
| | • dofetilide | |
| | • dronedarone | |
| | • flecainide | |
| | • ibutilide | |
| | • procainamide | |
| | • propafenone | |
| | • quinidine | |
| | • sotalol, d-sotalol | |


| <b>Medication Class</b> | Medicationa | Prohibition/restrictions |
|---|---|---|
| Anticholinergics | PROHIBITED • Centrally acting anticholinergics ○ biperiden ○ trihexiphenidyl | Centrally acting anticholinergic medications are prohibited throughout the treatment period. |
| | RESTRICTED o benztropine o oral diphenhydramine | <ul> <li>○ Benztropine (≤6 mg/day) is allowed for movement disorders</li> <li>○ Oral diphenhydramine is allowed at ≤50 mg per day for acute extrapyramidal symptoms</li> </ul> |
| | <ul> <li>UNRESTRICTED</li> <li>peripherally acting anticholinergics</li> <li>topical diphenhydramine</li> </ul> | Peripherally acting anticholinergic medications and topical diphenhydramine are allowed without restriction |
| Anticonvulsant and mood stabilizers | PROHIBITED carbamazepine lamotrigine lithium oxcarbazepine phenytoin valproate | Prohibited throughout the treatment period |
| Antidepressants | PROHIBITED amitriptyline citalopram clomipramine desipramine desvenlafaxine doxepin duloxetine escitalopram esketamine fluvoxamine fluoxetine imipramine ketamine mianserin mirtazapine | Prohibited throughout the treatment period |

| nefazadone nortriptyline sertraline trazodone trimipramine venlafaxine Antimanic agents PROHIBITED lithium valproate Antimicrobials, antifungals, and antimalarials PROHIBITED clarithromycin levofloxacin moxifloxacin pentamidine roxithromycin RESTRICTED artenimol/piperaquine azithromycin bedaquiline ciprofloxacin bedaquiline ciprofloxacin rottered but may be used during the course of the study to treat a bacterial infection (e.g., urinary tracinalisection, respiratory infection), post-Baseline at the discretion of the Investigator These restricted medications are only allowed under | Medication Class |
|---|---|
| sertraline trazodone trimipramine venlafaxine PROHIBITED lithium valproate Antimicrobials, antifiungals, and antimalarials PROHIBITED clarithromycin levofloxacin moxifloxacin pentamidine roxithromycin RESTRICTED artenimol/piperaquine azithromycin bedaquiline Prohibited throughout the treatment period | |
| trazodone trimipramine venlafaxine PROHIBITED lithium valproate Antimicrobials, antifungals, and antimalarials PROHIBITED clarithromycin levofloxacin pentamidine roxithromycin RESTRICTED artenimol/piperaquine azithromycin azithromycin azithromycin bedaquiline Prohibited throughout the treatment period | |
| trimipramine venlafaxine PROHIBITED lithium valproate Antimicrobials, antifungals, and antimalarials PROHIBITED clarithromycin levofloxacin moxifloxacin pentamidine roxithromycin RESTRICTED artenimol/piperaquine azithromycin azithromycin bedaquiline Prohibited throughout the treatment period | |
| Prohibited throughout the treatment period Prohibited throughout the treatment period | |
| Antimanic agents PROHIBITED Ithium valproate Antimicrobials, antifungals, and antimalarials clarithromycin levofloxacin moxifloxacin pentamidine roxithromycin RESTRICTED artenimol/piperaquine azithromycin bedaquiline Prohibited throughout the treatment period | |
| Antimicrobials, and antimalarials PROHIBITED clarithromycin levofloxacin moxifloxacin pentamidine roxithromycin RESTRICTED artenimol/piperaquine azithromycin bedaquiline Prohibited throughout the treatment period | |
| Antimicrobials, antifungals, and antimalarials PROHIBITED • clarithromycin • erythromycin • levofloxacin • moxifloxacin • pentamidine • roxithromycin RESTRICTED • artenimol/piperaquine • azithromycin • bedaquiline • valproate Prohibited throughout the treatment period | ıtimanic agents |
| Antimicrobials, antifungals, and antimalarials PROHIBITED • clarithromycin • levofloxacin • moxifloxacin • pentamidine • roxithromycin RESTRICTED • artenimol/piperaquine • azithromycin • bedaquiline Prohibited throughout the treatment period | |
| <ul> <li>clarithromycin</li> <li>erythromycin</li> <li>levofloxacin</li> <li>pentamidine</li> <li>roxithromycin</li> <li>RESTRICTED</li> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> </ul> <ul> <li>clarithromycin</li> <li>Prohibited but may be used during the course of the study to treat a bacterial infection (e.g., urinary traction, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | |
| <ul> <li>erythromycin</li> <li>levofloxacin</li> <li>moxifloxacin</li> <li>pentamidine</li> <li>roxithromycin</li> <li>RESTRICTED</li> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> <li>Prohibited but may be used during the course of the study to treat a bacterial infection (e.g., urinary trading infection, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | |
| <ul> <li>erythromycin</li> <li>levofloxacin</li> <li>moxifloxacin</li> <li>pentamidine</li> <li>roxithromycin</li> <li>RESTRICTED</li> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> <li>Prohibited but may be used during the course of the study to treat a bacterial infection (e.g., urinary trading infection, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | |
| <ul> <li>moxifloxacin</li> <li>pentamidine</li> <li>roxithromycin</li> <li>RESTRICTED</li> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> <li>Prohibited but may be used during the course of the study to treat a bacterial infection (e.g., urinary traction, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | imaiariais |
| <ul> <li>pentamidine</li> <li>roxithromycin</li> <li>RESTRICTED</li> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> <li>Prohibited but may be used during the course of the study to treat a bacterial infection (e.g., urinary traction, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | |
| <ul> <li>roxithromycin</li> <li>RESTRICTED <ul> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> </ul> </li> <li>Prohibited but may be used during the course of the study to treat a bacterial infection (e.g., urinary trading infection, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | |
| <ul> <li>RESTRICTED</li> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> <li>Prohibited but may be used during the course of the study to treat a bacterial infection (e.g., urinary traction, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | |
| <ul> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> <li>artenimol/piperaquine</li> <li>study to treat a bacterial infection (e.g., urinary traction, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | |
| <ul> <li>artenimol/piperaquine</li> <li>azithromycin</li> <li>bedaquiline</li> <li>study to treat a bacterial infection (e.g., urinary traction, respiratory infection), post-Baseline at the discretion of the Investigator</li> </ul> | |
| bedaquiline discretion of the Investigator The approximate density of the Investigator density of the Investigator The approximate density of the Investigator d | |
| The second standard and it settings are selected and and | |
| • These restricted medications are only allowed under | |
| - ciprojioxuciii | |
| • fluconazole the following conditions: | |
| • gemifloxacin • The subject has a Baseline ECG with a QTcF < 425 ms IF QRS duration is < 120 ms OR | |
| • norfloxacin • norfloxacin • The subject has a QTcF < 450 ms at Baseline IF | |
| • ofloxacin QRS duration ≥120 ms | |
| • telavancin | |
| telithromycin | |
| Antipsychotics other PROHIBITED Prohibited throughout the treatment period | |
| than pimavanserin All in class | an pimavanserin |
| Anxiolytics PROHIBITED Prohibited throughout the treatment period | ıxiolytics |
| • chlordiazepoxide | |
| • diazepam | |
| • flurazepam | |
| **RESTRICTED** • Mild sedation is allowed exceptionally for ECGs an | |
| • alprazolam blood draws during the study (e.g., alprazolam at a | |
| • lorazepam pediatric-appropriate dose per age, and the <u>lowest</u> | |
| • midazolam <u>dose</u> deemed necessary by the Investigator) just in | |

| Medication Class | Medicationa | Prohibition/restrictions |
|---|---|---|
| | <ul><li>oxazepam</li><li>temazepam</li><li>triazolam</li></ul> | cases when the subject's agitation/anxiety does not allow a safe and accurate measurement and the Investigator, with agreement from the caregiver, considers it safe and appropriate for the subject. • Short- or medium-acting benzodiazepine may be used for acute anxiety |
| | | <ul> <li>May not be used within 12 hours prior to an assessment visit</li> <li>Lorazepam, in doses according to age, may be used as a rescue medication for a maximum of 7 consecutive days. Reassessment and discussion with Medical Monitor is required if needed beyond 7 days.</li> <li>If lorazepam is not available, another benzodiazepine from the restricted list may be used</li> </ul> |
| Beta blockers | PROHIBITED • propranolol | Prohibited throughout the treatment period |
| Centrally-acting alpha-agonist hypotensive agents | PROHIBITED • clonidine | Prohibited throughout the treatment period |
| Centrally-acting alpha <sub>2A</sub> adrenergic receptor agonists | PROHIBITED • guanfacine | Prohibited throughout the treatment period |
| Hypnotics and sleeping agents | <ul><li>PROHIBITED</li><li>eszopiclone</li><li>zolpidem</li><li>zopiclone</li></ul> | Prohibited throughout the treatment period |
| | <ul><li>RESTRICTED</li><li>melatonin</li><li>ramelteon</li><li>zaleplon</li></ul> | May not be used within 12 hours of a cognitive assessment, and efforts should be made to limit agents to lowest dose for the shortest time needed. ○ Melatonin is allowed (≤5 mg/day) for insomnia |
| Non-stimulant<br>ADHD medications | **RESTRICTED * atomoxetine | Allowed if stable throughout the antecedent study and the dose is expected to remain the same throughout the duration of the study. |
| Opioids | PROHIBITED • methadone | Prohibited throughout the treatment period |
| Serotonin<br>antagonists | <ul><li>PROHIBITED</li><li>cyproheptadine</li></ul> | Prohibited throughout the treatment period |

| <b>Medication Class</b> | Medicationa | Prohibition/restrictions |
|---|---|---|
| Stimulants and<br>wake-promoting<br>agents | RESTRICTED amphetamine salts armodafinil lisdexamfetamine methylphenidate modafinil | Allowed if stable throughout the antecedent study and the dose is expected to remain the same throughout the duration of the study. |

Abbreviations: ADHD=attention-deficit hyperactivity disorder; ECG=electrocardiogram; QTcF=corrected QT interval using Fridericia's correction method; QRS=QRS interval on ECG; QT interval=QT interval on ECG


<sup>&</sup>lt;sup>a</sup> Medications within each class include but are not limited to the examples listed in this table.

# Appendix B Prohibited and Restricted Concomitant Medications: Inhibitors and Inducers of Cytochrome P450 Enzyme 3A4

The information presented here is intended to provide guidance and does not constitute an exhaustive list of strong CYP 3A4 enzyme (CYP3A4) inhibitors and inducers. Any questions should be discussed with the Medical Monitor or appropriate designee.

Subjects who require current treatment with a prohibited medication will be withdrawn from the study.

Subjects who have previously taken a prohibited medication during the study will be withdrawn from the study unless:

- the prohibited medication has been discontinued AND
- withdrawal from the study presents an unacceptable medical risk to the subject

The justification to allow the subject to continue in the study will be made by the Sponsor/Medical Monitor with medical input from the Investigator, and will be documented. If allowed to remain in the study, this will be reported as a major protocol deviation and not a waiver.

The metabolism of pimavanserin is affected by strong CYP3A4 inhibitors, resulting in an increase in  $C_{max}$  and AUC of approximately 3-fold.

Strong inhibitors of CYP3A4 are to be stopped at least <u>2 weeks or 5 half-lives</u> prior to investigational product administration, whichever is longer. Strong inducers of CYP3A4 are to be stopped <u>30 days or 5 half-lives</u> prior to investigational product administration, whichever is longer. Moderate inhibitors and inducers of CYP3A4 are allowed but should be used with caution.

| STRONG | grapefruit juice <sup>a</sup> | MODERATE | grapefruit juice <sup>a</sup> |
|---|---|---|---|
| INHIBITORS | boceprevir (Victrelis®) | INHIBITORS | amprenavir (Agenerase®) |
| | clarithromycin (Biaxin®) | | aprepitant (Emend®) |
| | cobicistat (part of Stribild®) | | atazanavir (Reyataz®) |
| | indinavir (Crixivan®) | | ciprofloxacin (Cipro®) |
| | itraconazole (Sporanox®) | | conivaptan (Vaprisol®) |
| | ketoconazole (Nizoral®) | | crizotinib |
| | lopinavir and ritonavir (Kaletra®) | | cyclosporine |
| | mibefradil (Posicor®) | | darunavir/ritonavir |
| | nefazodone (Serzone®) | | (Prezista®/Ritonavir) |
| | nelfinavir (Viracept®) | | diltiazem |
| | posaconazole (Noxafil®) | | dronedarone |
| | quinupristin (Synercid®) | | erythromycin (Erythrocin® |
| | ritonavir (Norvir®, part of Viekira | | Lactobionate) |
| | Pak <sup>TM</sup> ) | | fluconazole (Diflucan®) |


| | - combination treatments including ritonavir, such as: danoprevir and ritonavir elvitegravir and ritonavir indinavir and ritonavir lopinavir and ritonavir paritaprevir and ritonavir and ombitasvir (and/or dasabuvir) saquinavir and ritonavir tipranavir and ritonavir saquinavir (Invirase®) telaprevir (Incivek®) telithromycin (Ketek®) troleandomycin voriconazole (Vfend®) | | fluvoxamine (Luvox®) fosamprenavir (Lexiva®) imatinib (Gleevec®) isavuconazole tofisopam verapamil (Calan®) |
|---|---|---|---|
| STRONG<br>INDUCERS | apalutamide avasimibe carbamazepine (Tegretol®) enzalutamide ivosidenib lumacaftor mitotane phenytoin (Dilantin®) rifampin (Rifadin®, Rifadin® IV, Rimactane®) St. John's Wort | MODERATE<br>INDUCERS | bosentan (Tracleer®) cenobamate dabrafenib efavirenz (Sustiva®) etravirine (Intelence®) lorlatinib modafinil (Provigil®) nafcillin (Unipen®, Nallpen®) pexidartinib phenobarbital (Luminal®, Solfoton®) primidone sotorasib |

The effect of grapefruit juice varies widely among brands and is concentration-, dose-, and preparation-dependent. Studies have shown that it can be classified as a "strong CYP3A inhibitor" when a certain preparation was used (e.g., high dose, double strength) or as a "moderate CYP3A inhibitor" when another preparation was used (e.g., low dose, single strength). (FDA Drug Development and Drug Interactions http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/uc m093664.htm#classInhibit).

Appendix C Criteria for Identifying Potentially Clinically Important Laboratory Values

| Analyte | Conventional Unit | Low PCI Criteria | High PCI Criteria |
|---|---|---|---|
| Hematology (whole blood) | | | |
| Hemoglobin (Male) | g/dL | <11 | >17 |
| Hemoglobin (Female) | g/dL | <10 | >17 |
| Hematocrit (Both) | % | <30 | >50 |
| Leukocyte (White Blood Cell | $\times 10^3/\text{uL}$ | ≤2.8 | ≥15 |
| Count) | | | |
| Neutrophils | $\times 10^3/\text{uL}$ | ≤1.5 | No upper limit |
| Eosinophils | % | ≥10% | No lower limit |
| Platelet Count | $\times 10^3/\text{uL}$ | ≤75 | ≥700 |
| Chemistry (serum or plasma) | | | |
| ALT (SGPT) | U/L | No lower limit | ≥3 × ULN |
| AST (SGOT) | U/L | No lower limit | ≥3 × ULN |
| Gamma-Glutamyl Transferase | U/L | No lower limit | ≥3 ULN |
| (GGT) | | | |
| Lactate Dehydrogenase (LDH) | U/L | No lower limit | ≥3 × ULN |
| Alkaline Phosphatase | U/L | No lower limit | ≥3 × ULN |
| Total Bilirubin | mg/dL | No lower limit | ≥1.5 ULN |
| СРК | mg/dL | No lower limit | ≥3 ULN |
| BUN | mg/dL | No lower limit | ≥30.0 |
| Serum Creatinine | mg/dL | Not Applicable | >1.5 ULN |
| Sodium | mEq/L | ≤125 | ≥155 |
| Potassium | mEq/L | ≤3.0 | ≥5.5 |
| Calcium, total | mg/dL | <8.0 | >11.0 |
| Chloride | mEq/L | ≤85 | ≥120 |
| Phosphorous, inorganic | mg/dL | ≤1.0 mg/dL | ≥4.5 mg/dL |
| Magnesium | mEq/L | ≤0.7 mEq/L | ≥5.0 mEq/L |
| Uric acid | mg/dL | No lower limit | ≥8.5 |
| Albumin | g/dL | ≤2.6 | ≥6.0 |
| Total Protein | g/dL | ≤5.0 | ≥10.0 |
| Glucose (random) | mg/dL | ≤45.1 | ≥115.0 |
| Hb1Ac | % | No lower limit | ≥7% |
| Total Cholesterol, Fasting | mg/dL | No lower limit | ≥240 mg/dL |
| Urinalysis | | | |
| Blood (occult blood) | | Not Applicable | ≥ Moderate |
| Protein | mg/dL | Not Applicable | ≥100 mg/dL |
| Glucose | mg/dL | Not Applicable | ≥500 mg/dL |

Abbreviations: ALT (SGPT)=alanine aminotransferase (serum glutamic-pyruvic transaminase);

AST (SGOT)=aspartate aminotransferase (serum glutamic-oxaloacetic transaminase); BUN=blood urea nitrogen; CPK=creatine phosphokinase;  $HbA_{1c}$ =glycosylated hemoglobin; PCI=potentially clinically important; ULN=upper limit of normal.


Appendix D Criteria for Potentially Clinically Important ECG Values

| ECG Parameter | High PCI Criteria |
|----------------------------|-------------------|
| QRS Interval | ≥120 ms |
| PR Interval | ≥220 ms |
| QTcB | >500 ms |
| QTcF | >500 ms |
| QTcB: change from baseline | >60 ms |
| QTcF: change from baseline | >60 ms |

Abbreviations: ECG=electrocardiogram; PCI=potentially clinically important; PR interval=PR interval on ECG; QRS interval=QRS interval on ECG; QTcB=corrected QT interval using Bazett's correction method; QTcF=corrected QT interval using Fridericia's correction method; QRS interval=QRS interval on ECG.

Study: ACP-103-070 Final Version: 2.0 Clinical Study Protocol Amendment 3-Consolidated Date: 29 February 2024

Appendix E Criteria for Identifying Additional ECG Measurements of Potential Clinical Relevance. To be Used for Medical Monitoring Purposes

| | Variable | Criterion Value <sup>a</sup> | Change Relative to<br>Baseline |
|---|---|---|---|
| Rate | | | |
| | Tachycardia | ≥120 bpm | increase of ≥15 bpm |
| | Bradycardia | ≤50 bpm | decrease of ≥15 bpm |
| Rhythm | | | |
| | Sinus tachycardia <sup>b</sup> | ≥120 bpm | increase of ≥15 bpm |
| | Sinus bradycardia <sup>c</sup> | ≤50 bpm | decrease of ≥15 bpm |
| | Supraventricular premature beat | all | not present - present |
| | Ventricular premature beat | all | not present - present |
| | Supraventricular tachycardia | all | not present - present |
| | Ventricular tachycardia | all | not present - present |
| | Atrial fibrillation | all | not present - present |
| | Atrial flutter | all | not present - present |
| Conduction | | | |
| | 1st atrioventricular block | PR <u>≥</u> 0.20 second | increase of ≥0.05 second |
| | 2nd atrioventricular block | all | not present - present |
| | 3rd atrioventricular block | all | not present - present |
| | Left bundle-branch block | all | not present - present |
| | Right bundle-branch block | all | not present - present |
| | Pre-excitation syndrome | all | not present - present |
| | Other intraventricular conduction block | QRS ≥0.12 second | increase of 0.02 second |
| Infarction | | | |
| | Acute or subacute | all | not present - present |
| | Old | all | not present - present |
| ST/T Morphological | | | ≥12 weeks post trial entry |
| | Myocardial Ischemia | all | not present - present |
| | Symmetrical T-wave inversion | all | not present - present |
| | Increase in QTc | QTc | |
| | | ≥450 ms (males) | ≥10% increase |
| | | ≥470 ms (females) | |

In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

b No current diagnosis of supraventricular tachycardia, ventricular tachycardia, atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>c</sup> No current diagnosis of atrial fibrillation, atrial flutter, or other rhythm abnormality.

Appendix F Criteria for Potentially Clinically Important Vital Signs

| | | Criteria | | |
|---|---|---|---|---|
| Vital Sign Parameter | Unit | Observed Value | And/Or | Change Relative to<br>Baseline |
| Systolic blood pressure (supine or sitting) | mmHg | ≥140 | And | Increase of ≥20 |
| | | ≤70 | And | Decrease of ≥20 |
| Diastolic blood pressure (supine or sitting) | mmHg | ≥90 | And | Increase of ≥15 |
| | | ≤50 | And | Decrease of ≥15 |
| Pulse (supine or sitting) | bpm | ≥120 | And | Increase of ≥15 |
| | | ≤50 | And | Decrease of ≥15 |
| Weight | kg | Not Applica | able | Increase of ≥7% |
| | | | | Decrease of ≥7% |

# **Appendix G** Syncope Adverse Event Questions




# Appendix H Somnolence Adverse Event Questions

| • | CCI |
|---|-----|
| ı | |
| • | |